CLINICAL TRIAL: NCT03583697
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Safety and Efficacy of BMN 111 in Infants and Young Children With Achondroplasia, Age 0 to < 60 Months
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of BMN 111 in Infants and Young Children With Achondroplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111-206; 2016-003826-18 (EudraCT Number)
Record Dates: First submitted 2018-06-14; First posted 2018-07-11 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Achondroplasia
Keywords: Dwarfism; Bone Diseases; Bone Diseases, Developmental; ACH; Natriuretic Peptide, C-Type; Musculoskeletal Diseases; Natriuretic Agents; Physiological Effect of Drugs; Skeletal Dysplasias; Genetic Diseases, Inborn; Osteochondrodysplasias
MeSH Terms: conditions — Achondroplasia; Dwarfism; Bone Diseases; Bone Diseases, Developmental; Musculoskeletal Diseases; Genetic Diseases, Inborn; Osteochondrodysplasias | interventions — vosoritide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active BMN111 (Experimental): Subcutaneous injection of 15 μg/kg/day and/or 30 μg/kg/day of BMN111 daily.
  Interventions: Drug: BMN 111
- Placebo (Placebo Comparator): Daily subcutaneous injection of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMN 111 — Subcutaneous injection of 15 μg/kg/day and/or 30 μg/kg/day of BMN 111 daily, subject to adjustment per protocol
  Other Names: Vosoritide; Modified recombinant human C-type natriuretic peptide
  Arms: Active BMN111
Drug: Placebo — Subcutaneous injection of 15 μg/kg of placebo daily, Subject to adjustment per protocol
  Arms: Placebo

SUMMARY:
Study 111-206 is a Phase 2 randomized, double-blind, placebo-controlled clinical trial of BMN 111 in infants and young children with a diagnosis of achondroplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of achondroplasia (ACH), confirmed by genetic testing. If subjects had previous genetic testing, subjects must have a lab report from a certified laboratory with the study specific mutation documented.
2. Age 0 to < 60 months, at study entry (Day 1)
3. Cohort 1 and 2 subjects must have at least a 6-month period of pretreatment growth assessment in Study 111 901 immediately before screening, and have one documented measurement of height/body length a minimum of 6 months prior to the screening visit for 111-206. Cohort 3 subjects must have a minimum of 3 months of observation prior to treatment. This observational period can be obtained either (1) via prior enrollment in Study 111-901 or (2) via enrollment in this Study 111 206 for a minimum of 3 months of non-treatment observation prior to commencement of treatment.
4. Parent(s) or guardian(s) (and the subjects themselves, if required by local regulations or ethics committee) are willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to performance of any research-related procedure
5. Willing and able to perform all study procedures as physically possible
6. Parent(s) or caregiver(s) are willing to administer daily injections to the subjects and complete the required training

Exclusion Criteria:

1. Have hypochondroplasia or short-stature condition other than achondroplasia (e.g., trisomy 21, pseudoachondroplasia, etc.)
2. Subject weighs < 5.0 kg (Cohort 1 and 2) or < 4.0 kg (Cohort 3)
3. Have any of the following:

   * Hypothyroidism or hyperthyroidism
   * Insulin-requiring diabetes mellitus
   * Autoimmune inflammatory disease (including celiac disease, systemic lupus erythematosus, juvenile dermatomyositis, scleroderma, etc.)
   * Inflammatory bowel disease
   * Autonomic neuropathy
4. Have a history of any of the following:

   * Renal insufficiency defined as serum creatinine > 2 mg/dL
   * Chronic anemia or Hgb <10.0 g/dL (based on screening clinical laboratory testing)
   * Baseline systolic blood pressure (BP) below age and gender specified normal range or recurrent symptomatic hypotension (defined as episodes of low BP generally accompanied by symptoms e.g., dizziness, fainting) or recurrent symptomatic orthostatic hypotension
   * Cardiac or vascular disease, including the following

     * Cardiac dysfunction (abnormal echocardiogram determined to be clinically significant by principal investigator PI and medical monitor) at Screening Visit
     * Hypertrophic cardiomyopathy
     * Pulmonary hypertension
     * Congenital heart disease with ongoing cardiac dysfunction
     * Cerebrovascular disease
     * Aortic insufficiency or other clinically significant valvular dysfunction
     * Clinically significant atrial or ventricular arrhythmias
5. Have a clinically significant finding or arrhythmia that indicates abnormal cardiac function or conduction or Fridericia's corrected QT interval (QTc-F) >450 msec on screening ECG
6. Have evidence of cervicomedullary compression (CMC) likely to require surgical intervention within 60 days of Screening as determined by the Investigator based on the following assessments

   * Physical exam (e.g., neurologic findings of clonus, opisthotonus, exaggerated reflexes, dilated facial veins)
   * Polysomnography (e.g., severe central sleep apnea)
   * MRI indicating presence of severe CMC or spinal cord damage
7. Have an unstable medical condition likely to require surgical intervention in the next 6 months, or planned spine or long-bone surgery (i.e., surgery involving significant disruption of bone cortex) during the study period
8. Have documented uncorrected Vitamin D deficiency: 25(OH)D <=15 ng/mL (37.5 nmol/L)
9. Require any other investigational product prior to completion of the study period
10. Have received another investigational product or investigational medical device within 30 days prior to the Screening visit
11. Have used any other investigational product or investigational medical device for the treatment of achondroplasia or short stature at any time
12. Require current chronic therapy with antihypertensive medication or any medication that, in the investigator's judgment, may compromise the safety or ability of the subject to participate in this clinical study (Table 9.3.5.1)
13. Have been treated with growth hormone, insulin-like growth factor 1 (IGF-1), or anabolic steroids in the 6 months prior to screening, or long-term treatment (>3 months) at any time
14. Have had regular long-term treatment (> 1 month) with oral corticosteroids (low-dose ongoing inhaled steroid for asthma, or intranasal steroids, are acceptable) in the 12 months prior to screening
15. Have ever had cervicomedullary decompression surgery (Cohorts 2 and 3 only), spine or long-bone surgery (i.e., surgery involving disruption of bone cortex) or have ever had bone-related surgery with chronic complications

    NOTE: Subjects with prior cervicomedullary decompression may be allowed into Cohort 1 only after discussion and agreement with Medical Monitor.
16. Have ever had limb-lengthening surgery or plan to have limb-lengthening surgery during the study period
17. Have had a fracture of the long bones or spine within 6 months prior to screening
18. Have aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or total bilirubin greater than upper limit of normal (ULN) at screening (except for subjects with a known history of Gilberts or newborns entering screening in Cohort 3)
19. Have evidence of severe untreated sleep apnea; or have newly initiated sleep apnea treatment (eg, Continuous positive airway pressure (CPAP) or sleep apnea-mitigating surgery) in the 2 months prior to screening
20. Have current malignancy, history of malignancy, or currently under work-up for suspected malignancy
21. Have known hypersensitivity to BMN 111 or its excipients
22. Have a history of hip surgery or severe hip dysplasia
23. Have a history of clinically significant hip injury in the 30 days prior to screening
24. Have a history of slipped capital femoral epiphysis or avascular necrosis of the femoral head
25. Have abnormal findings on baseline clinical hip exam or imaging assessments that are determined to be clinically significant as determined by the Investigator
26. Have a condition or circumstance that, in the view of the Investigator, places the subject at high risk for poor treatment compliance or for not completing the study
27. Have any concurrent disease or condition that, in the view of the Investigator, would interfere with study participation or safety evaluations, for any reason

Inclusion Criteria for Cohort 3 Observation Period

1. Parent(s) or guardian(s) willing and able to provide signed informed consent after the nature of the study has been explained and prior to performance of any research-related procedure. Also, willing and able to provide written assent (if applicable) after the nature of the study has been explained and prior to performance of any research-related procedure.
2. Birth to <= 3 months of age at study entry.
3. Have ACH, documented by genetic testing
4. Are willing and able to perform all study procedures as physically possible

Exclusion Criteria for Cohort 3 Observation Period

1. Have hypochondroplasia or short stature condition other than ACH (e.g., trisomy 21, pseudoachondroplasia)
2. Have any of the following disorders:

   * Hypothyroidism
   * Insulin-requiring diabetes mellitus
   * Autoimmune inflammatory disease (including celiac disease, lupus (SLE), juvenile dermatomyositis, scleroderma, and others)
   * Inflammatory bowel disease
   * Autonomic neuropathy
3. Have an unstable clinical condition likely to lead to intervention during the course of the study, including progressive cervical medullary compression
4. Have a history of any of the following:

   * Renal insufficiency
   * Anemia
5. Have a history of cardiac or vascular disease, including the following:

   * Cardiac dysfunction
   * Hypertrophic cardiomyopathy
   * Congenital heart disease
   * Cerebrovascular disease, aortic insufficiency
   * Clinically significant atrial or ventricular arrhythmias
6. Current treatment with antihypertensive medications, angiotensin-converting enzyme (ACE) inhibitors, angiotensin II receptor blockers, diuretics, beta-blockers, calcium-channel blockers, cardiac glycosides, systemic anticholinergic agents, any medication that may impair or enhance compensatory tachycardia, drugs known to alter renal function that is expected to continue for the duration of the study
7. Have had regular long-term treatment (> 1 month) with oral corticosteroids (low-dose ongoing inhaled steroid for asthma is acceptable) in the previous 3 month
8. Concomitant medication that prolongs the QT/QTc interval within 14 days or 5 half-lives, whichever is longer, before the Screening visit
9. Have used any other investigational product or investigational medical device for the treatment of ACH or short stature
10. Planned or expected bone-related surgery (ie. surgery involving disruption of bone cortex), during the study period.
11. Planned or expected to have limb-lengthening surgery during the study period.
12. Have any condition that, in the view of the Investigator, places the subject at high risk of poor compliance with the visit schedule or of not completing the study.
13. Concurrent disease or condition that, in the view of the Investigator, would interfere with study participation

Max Age: 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (16):
- United States (9):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Emory University, Decatur, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin, Children's Hospital, Milwaukee, Wisconsin
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Murdoch Children's Research Institute, Parkville, Victoria
- Japan (3):
  - Osaka University Hospital, Osaka
  - Saitama Children's Medical Center, Saitama
  - Tokushima University Hospital, Tokushima
- United Kingdom (2):
  - Guy's and St. Thomas NHS Foundation Trust Evelina Children's Hospital, London
  - Sheffield Children's NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qi Y, Chan ML, Mould DR, Larimore K, Fisheleva E, Cherukuri A, Day J, Savarirayan R, Irving M, Bacino CA, Hoover-Fong J, Ozono K, Mohnike K, Wilcox WR, Bober MB, Henshaw J. Development of a Weight-Band Dosing Approach for Vosoritide in Children with Achondroplasia Using a Population Pharmacokinetic Model. Clin Pharmacokinet. 2024 May;63(5):707-719. doi: 10.1007/s40262-024-01371-6. Epub 2024 Apr 23. PMID 38649657
- [Derived] Savarirayan R, Wilcox WR, Harmatz P, Phillips J 3rd, Polgreen LE, Tofts L, Ozono K, Arundel P, Irving M, Bacino CA, Basel D, Bober MB, Charrow J, Mochizuki H, Kotani Y, Saal HM, Army C, Jeha G, Qi Y, Han L, Fisheleva E, Huntsman-Labed A, Day J. Vosoritide therapy in children with achondroplasia aged 3-59 months: a multinational, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Child Adolesc Health. 2024 Jan;8(1):40-50. doi: 10.1016/S2352-4642(23)00265-1. Epub 2023 Nov 18. PMID 37984383
- See also: NIH Genetics Home Reference related topics: Achondroplasia — https://ghr.nlm.nih.gov/condition/achondroplasia
- See also: Description NIH Genetic and Rare Diseases Information Center resources: Achondroplasia — https://rarediseases.info.nih.gov/diseases/8173/achondroplasia
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center study conducted by 16 principal investigators at 16 study centers in four countries (United States, Australia, United Kingdom and Japan).
Pre-assignment Details: A total of 75 participants (full analysis set [FAS]) were enrolled into the study, of which 11 participants were enrolled to receive vosoritide (sentinel participants). 64 participants were blinded and randomized to receive vosoritide or placebo (32 randomized for vosoritide and 32 for placebo), which constituted the FAS (randomized).
Groups:
- Sentinel: Cohort 1 Sentinel: Participants stratified by age >= 24 to < 60 months, received vosoritide 15 µg/kg/day single daily subcutaneous injection (n=4)
  Cohort 2 Sentinel: Participants stratified by age >= 6 to < 24 months, received vosoritide 15 µg/kg/day & 30 µg/ kg/day single daily subcutaneous injection (n=4)
  Cohort 3 Sentinel: Participants stratified by age 0 to < 6 months, received vosoritide 30 µg/kg/day single daily subcutaneous injection (n=3)
- Randomized Vosoritide: Cohort 1: Participants stratified by age >= 24 to < 60 months, received vosoritide 15 µg/kg/day single daily subcutaneous injection (n=15)
  Cohort 2: Participants stratified by age >= 6 to < 24 months, received vosoritide 15 µg/kg/day & 30 µg/kg/day single daily subcutaneous injection (n=8)
  Cohort 3: Participants stratified by age 0 to < 6 months, received vosoritide 30 µg/kg/day single daily subcutaneous injection (n=9)
- Randomized Placebo: Cohort 1: Participants stratified by age >= 24 to < 60 months, received placebo single daily subcutaneous injection (n=16)
  Cohort 2: Participants stratified by age >= 6 to < 24 months, received placebo single daily subcutaneous injection (n=8)
  Cohort 3: Participants stratified by age 0 to < 6 months, received placebo single daily subcutaneous injection (n=8)
Period: Overall Study
Arm/Group | Sentinel | Randomized Vosoritide | Randomized Placebo
Started | 11 | 32 | 32
Cohort 1: Age >= 24 to < 60 Months | 4 | 15 | 16
Cohort 2: Age >= 6 to < 24 Months | 4 | 8 | 8
Cohort 3: Age 0 to < 6 Months | 3 | 9 | 8
Completed | 11 | 31 | 31
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — AE of sudden infant death syndrome, not related | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: FAS Population: The Full Analysis Set (FAS) was defined according to the intent-to-treat principle and included all enrolled sentinel and randomized participants with a signed informed consent.
Groups:
- Sentinel: Cohort 1 Sentinel: Participants stratified by age >= 24 to < 60 months, received vosoritide 15 µg/kg/day single daily subcutaneous injection (n=4)
  Cohort 2 Sentinel: Participants stratified by age >= 6 to < 24 months, received vosoritide 15 µg/kg/day & 30 µg/kg/day single daily subcutaneous injection (n=4)
  Cohort 3 Sentinel: Participants stratified by age 0 to < 6 months, received vosoritide 30 µg/kg/day single daily subcutaneous injection (n=3)
- Total: Total of all reporting groups
Arm/Group | Sentinel | Randomized Vosoritide | Randomized Placebo | Total
Number analyzed (Participants) | 11 | 32 | 32 | 75
Age, Continuous [Mean (Standard Deviation); unit: Months] — Age at Screening, months
  Months | 23.4 (21.0) | 23.0 (16.9) | 26.5 (19.3) | 24.5 (18.4)
Age, Continuous [Mean (Standard Deviation); unit: Months] — Age on Day 1, months.
  Months | 24.71 (20.79) | 24.39 (16.83) | 27.82 (19.25) | 25.90 (18.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 15 | 19 | 37
  Male | 8 | 17 | 13 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3 | 6
  Not Hispanic or Latino | 11 | 29 | 29 | 69
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Full analysis population (FAS).
  Participants
    White | 8 | 21 | 25 | 54
    Asian-Other | 1 | 6 | 2 | 9
    Asian-Japanese | 0 | 4 | 4 | 8
    Multiple | 2 | 1 | 0 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
Weight [Mean (Standard Deviation); unit: Kg] | 10.12 (3.70) | 10.20 (3.83) | 10.55 (4.31) | 10.34 (3.98)
Weight Z-Score [Mean (Standard Deviation); unit: Z-Score] — The weight Z-score represents the participant's weight converted to an age and sex appropriate standard deviation score (SDS) by comparison with an average stature reference population. The weight Z-score of 0 represents the mean weight for age and sex of the reference population. A positive weight Z-score means weight is above the mean weight for the average stature population of the same sex and age and a negative weight Z-Score means weight is below the mean weight for the average stature population of the same sex and age.
  Z-Score | -1.41 (0.73) | -1.49 (1.26) | -1.59 (1.44) | -1.52 (1.27)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI).
  For height used for BMI calculation, participants aged < 24 months, body length takes precedence over standing height.
  Participants aged < 24 months at baseline and >= 24 months at Week 52, body length takes precedence.
  kg/m^2 | 20.06 (1.87) | 19.48 (2.45) | 20.14 (2.39) | 19.85 (2.34)
BMI Z-Score [Mean (Standard Deviation); unit: Z-Score] — The body mass index (BMI) Z-score represents the participant's BMI converted to an age and sex appropriate standard deviation score (SDS) by comparison with an average stature reference population. The weight Z-score of 0 represents the mean BMI for age and sex of the reference population. A positive BMI Z-score means BMI is above the mean BMI for the average stature population of the same sex and age and a negative BMI Z-Score means BMI is below the mean BMI for the average stature population of the same sex and age. Population: BMI Z-Scores were derived only for participants aged 24 months or older. Hence, participants in Cohort 2 (n=Sentinel 4, Vosoritide 8, Placebo 8) and Cohort 3 (n=Sentinel 3, Vosoritide 9, Placebo 8) were are not included.
  Z-Score
    number analyzed (Participants) | 4 | 15 | 16 | 35
    (all) | 2.79 (0.98) | 2.52 (1.15) | 2.77 (0.75) | 2.67 (0.94)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) by Severity Grade and Study Drug Treatment-emergent Adverse Events (TEAEs)
Description: A treatment-emergent Adverse Events (TEAE) is any Adverse Events that newly appeared, increased in frequency or worsened in severity following initiation of study drug administration. A severity grade was defined by the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. As per CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to AE.
  Safety Population includes all sentinel and randomized participants in the FAS who received at least one dose of vosoritide or placebo in this study.
  Serious adverse event (SAE)
Time Frame: Up to Week 56 (Safety Follow-Up +/-7d)
Population: Safety Population: The Safety Population was a subset of the FAS who received at least one dose of vosoritide or placebo in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sentinel | Randomized Vosoritide | Randomized Placebo
Number analyzed (Participants) | 11 | 32 | 32
Participants
  Participants with any AE | 11 | 32 | 32
  Participants with any SAE | 0 | 3 | 6
  Participants with any treatment-related AE | 8 | 29 | 17
  Participants with any treatment-related SAEs | 0 | 0 | 0
  Participants with any AE of CTCAE grade >=3 | 0 | 2 | 3
  Participants who died | 0 | 1 | 0

2. Primary Outcome: Change From Baseline in Height Z-score at Week 52.
Description: Z-Scores were derived using age-sex specific reference data (means and SDS) for average stature children per the Centers for Disease Control and Prevention. A height Z score of 0 would indicate that the subject's height is equal to the mean height for the average stature population of the same sex and age. A positive height Z score indicates that the subjects height is above the mean height for the average stature population of the same sex and age, whilst a negative height Z score indicates that the subjects height is below the mean height for the average stature population of the same sex and age. To conclude if the height Z score increases then this means the height deficit has decreased.
  standard deviation score (SDS).
  The primary efficacy analysis population was the subset of randomized participants in the FAS.
Time Frame: Baseline to Week 52
Population: FAS & FAS (randomized) population:The FAS (randomized) was a subset of the FAS, which included 64 participants who were randomized to study treatment (32 participants randomized to vosoritide & 32 participants randomized to placebo).
  This is model-based analysis, it is true that the participants analyzed for placebo FAS & FAS (randomized) are the same, but participants analyzed for vosoritide arm FAS & FAS(randomized) are different, that's why the model-based results for placebo are different
Measure: Least Squares Mean (95% Confidence Interval); unit: Z-score
Groups:
- All Vosoritide: All Vosoritide : 11 sentinel + 32 randomized participants who received vosoritide 15 µg/kg/day or 30 µg/kg/day, single daily subcutaneous injection.
- Placebo: Placebo: Participants who received placebo single daily subcutaneous injection.
Arm/Group | Randomized Vosoritide | Randomized Placebo | All Vosoritide | Placebo
Number analyzed (Participants) | 32 | 32 | 43 | 32
Z-score | -0.06 [-0.26 to 0.15] | -0.31 [-0.48 to -0.13] | 0.01 [-0.15 to 0.17] | -0.30 [-0.47 to -0.13]
Statistical Analysis 1: Comparison: Randomized Vosoritide vs Randomized Placebo; Z-Scores were derived using age-sex specific reference data (means and SDs) for average stature children per the Centers for Disease Control and Prevention. Participants aged < 24 months, body length takes precedence over standing height. Participants aged < 24 months at baseline and >= 24 months at Week 52, body length takes precedence. Difference in least squares (LS) means were obtained from an analysis of covariance model; Test type: Superiority; Least Square Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.02 to 0.53]
Statistical Analysis 2: Comparison: All Vosoritide vs Placebo; Z-Scores were derived using age-sex specific reference data (means and SDs) for average stature children per the Centers for Disease Control and Prevention. Participants aged < 24 months, body length takes precedence over standing height. Participants aged < 24 months at baseline and >= 24 months at Week 52, body length takes precedence. Difference in LS means were obtained from an analysis of covariance model; Test type: Superiority; Least Square Mean Difference (Net) = 0.3, 95% CI 2-sided [0.07 to 0.54]

3. Secondary Outcome: Change From Baseline in Height at Week 52
Description: As a general rule, standing height/sitting height was used if participants were aged >= 24 months at baseline. Body length/crown to rump was used if participants were aged < 24 months at baseline. If body length was not measured and standing height was available, standing height was used.
Time Frame: Baseline to Week 52
Population: FAS (randomized) Population and FAS population.
  This is model-based analysis, it is true that the participants analyzed for placebo FAS & FAS (randomized) are the same, but participants analyzed for vosoritide arm FAS & FAS (randomized) are different, that's why the model-based results for placebo are different.
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Arm/Group | Randomized Vosoritide | Randomized Placebo | All Vosoritide | Placebo
Number analyzed (Participants) | 32 | 32 | 43 | 32
cm | 8.15 [7.55 to 8.75] | 7.38 [6.87 to 7.89] | 8.41 [7.93 to 8.89] | 7.45 [6.95 to 7.95]
Statistical Analysis 1: Comparison: Randomized Vosoritide vs Randomized Placebo; Difference in LS means were obtained from an analysis of covariance model; Test type: Superiority; Least Square Mean Difference (Net) = 0.77, 95% CI 2-sided [-0.02 to 1.56]
Statistical Analysis 2: Comparison: All Vosoritide vs Placebo; Difference in LS means were obtained from an analysis of covariance model; Test type: Superiority; Least Square Mean Difference (Net) = 0.96, 95% CI 2-sided [0.26 to 1.66]

4. Secondary Outcome: Change From Baseline in Annualized Growth Velocity (AGV) at Week 52
Description: AGV was derived over 12-month intervals starting from the baseline visit. Annualized growth velocity (AGV) = Standing Height at Date 2 - Standing Height at Date 1/Interval Length (Days) x 365.25.
  Difference in LS means were obtained from an analysis of covariance model.
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/year
Arm/Group | Randomized Vosoritide | Randomized Placebo | All Vosoritide | Placebo
Number analyzed (Participants) | 32 | 32 | 43 | 32
cm/year | -2.17 [-2.76 to -1.58] | -2.95 [-3.45 to -2.45] | -2.41 [-2.88 to -1.94] | -3.32 [-3.81 to -2.84]
Statistical Analysis 1: Comparison: Randomized Vosoritide vs Randomized Placebo; Test type: Superiority; Least Square Mean Difference (Net) = 0.78, 95% CI 2-sided [0.02 to 1.54]
Statistical Analysis 2: Comparison: All Vosoritide vs Placebo; Difference in LS means were obtained from an analysis of covariance model; Test type: Superiority; Least Square Mean Difference (Net) = 0.92, 95% CI 2-sided [0.24 to 1.59]

5. Secondary Outcome: Change From Baseline in Upper to Lower Body Segment Ratio at Week 52
Description: Upper to Lower Body ratio=Sitting Height / (Standing Height - Sitting Height).
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Randomized Vosoritide | Randomized Placebo | All Vosoritide | Placebo
Number analyzed (Participants) | 32 | 32 | 43 | 32
Ratio | -0.20 [-0.28 to -0.13] | -0.13 [-0.21 to -0.06] | -0.19 [-0.25 to -0.13] | -0.13 [-0.20 to -0.06]
Statistical Analysis 1: Comparison: Randomized Vosoritide vs Randomized Placebo; Difference in LS means were obtained from an analysis of covariance model; Test type: Superiority; Least Square Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.17 to 0.04]
Statistical Analysis 2: Comparison: All Vosoritide vs Placebo; Difference in LS means were obtained from an analysis of covariance model; Test type: Superiority; Least Square Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.15 to 0.03]

6. Secondary Outcome: Change From Baseline in Other Growth Measures (Upper Body Length, Head Circumference, Arm Span, Upper Arm Length, Lower Arm Length, Lower Body Length, Upper Leg Length, Knee to Heel Length, and Tibial Length) at Week 52
Description: Change from baseline in other growth measures (upper body length, head circumference, arm span, upper arm length, lower arm (Forearm) length, Lower Body Length, Upper Leg Length (Thigh), knee to heel length, and tibial length) at Week 52.
  Participants aged <24 months, body length and crown to rump length take precedence over standing height and sitting height. Participants aged <24 months at baseline and >=24 months at Week 52, body length and crown to rump length take precedence.
Time Frame: Baseline to Week 52
Population: FAS population.
  Change from baseline was based on the participants with available measurements at both time points. Baseline is defined as Day 1 or screening if a Day 1 measurement is not available.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Cohort 1: Placebo: Cohort 1 Placebo: Participants stratified by age >= 24 to < 60 months, received placebo single daily subcutaneous injection.
- Cohort 1: Vosoritide: Cohort 1 Vosoritide: Participants stratified by age >= 24 to < 60 months, received vosoritide 15 µg/kg/day single daily subcutaneous injection.
- Cohort 2: Placebo: Cohort 2 Placebo: Participants stratified by age >= 6 to < 24 months, received placebo single daily subcutaneous injection.
- Cohort 2: Vosoritide: Cohort 2 Vosoritide: Participants stratified by age >= 6 to < 24 months, received vosoritide 15 µg/kg/day & 30 µg/kg/day single daily subcutaneous injection.
- Cohort 3: Placebo: Cohort 3 Placebo: Participants stratified by age 0 to < 6 months, received placebo single daily subcutaneous injection.
- Cohort 3: Vosoritide: Cohort 3 Vosoritide: Participants stratified by age 0 to < 6 months, received vosoritide 30 µg/kg/day single daily subcutaneous injection.
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide | Cohort 3: Placebo | Cohort 3: Vosoritide
Number analyzed (Participants) | 16 | 19 | 7 | 12 | 8 | 11
cm
  Upper body length | 3.04 (1.52) | 3.54 (1.81) | 5.45 (1.75) | 5.20 (1.50) | 6.58 (0.99) | 6.75 (0.86)
  Head Circumference: number analyzed (Participants) | 16 | 19 | 7 | 11 | 8 | 11
  Head Circumference | 0.68 (0.66) | 0.74 (0.49) | 2.29 (1.28) | 3.10 (1.45) | 5.35 (0.71) | 6.29 (0.81)
  Arm Span: number analyzed (Participants) | 16 | 19 | 7 | 10 | 8 | 10
  Arm Span | 4.86 (1.99) | 5.82 (3.65) | 7.13 (1.59) | 7.22 (1.45) | 8.22 (1.93) | 8.99 (4.77)
  Upper Arm Length: number analyzed (Participants) | 16 | 19 | 7 | 11 | 8 | 11
  Upper Arm Length | 1.02 (1.13) | 0.77 (0.96) | 1.08 (0.93) | 1.44 (1.26) | 1.95 (1.23) | 1.44 (1.33)
  Lower Arm (Forearm) Length: number analyzed (Participants) | 16 | 19 | 7 | 10 | 8 | 11
  Lower Arm (Forearm) Length | 0.49 (0.96) | 0.79 (0.90) | 1.78 (0.44) | 1.57 (0.98) | 1.66 (0.82) | 1.49 (0.79)
  Lower Body Length | 2.41 (1.31) | 2.89 (1.99) | 2.39 (1.27) | 3.79 (1.56) | 3.86 (1.55) | 4.41 (1.53)
  Upper Leg Length (Thigh): number analyzed (Participants) | 16 | 19 | 7 | 10 | 8 | 11
  Upper Leg Length (Thigh) | 0.82 (1.75) | 1.55 (1.46) | 0.38 (1.71) | 1.10 (1.42) | 1.98 (2.21) | 1.93 (1.65)
  Knee to Heel Length: number analyzed (Participants) | 16 | 19 | 7 | 11 | 8 | 11
  Knee to Heel Length | 1.52 (0.76) | 2.21 (0.67) | 2.70 (0.75) | 2.29 (1.91) | 2.93 (0.68) | 3.12 (0.85)
  Tibial Length: number analyzed (Participants) | 16 | 19 | 7 | 11 | 8 | 11
  Tibial Length | 0.85 (0.69) | 1.16 (1.35) | 1.97 (1.49) | 1.99 (0.80) | 1.83 (0.88) | 1.39 (0.77)

7. Secondary Outcome: Change From Baseline in Other Body Proportion Ratios (Arm Span to Height Ratio, Upper Arm Length to Lower Arm [Forearm] Length Ratio, Upper Leg Length [Thigh] to Knee to Heel Length Ratio, and Upper Leg Length (Thigh) to Tibial Length Ratio) at Week 52
Description: For Height: subjects aged < 24 months, body length takes precedence over standing height. Subjects aged < 24 months at baseline and >= 24 months at Week 52, body length takes precedence.
Time Frame: Baseline to Week 52
Population: FAS population.
  Change from baseline was based on the subjects with available measurements at both time points. Baseline is defined as Day 1 or screening if a Day 1 measurement is not available
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide | Cohort 3: Placebo | Cohort 3: Vosoritide
Number analyzed (Participants) | 16 | 19 | 7 | 10 | 8 | 11
Ratio
  Upper Arm Length to Lower Arm(Forearm)Length Ratio | 0.05 (0.15) | 0.00 (0.12) | -0.09 (0.06) | 0.01 (0.10) | 0.02 (0.11) | -0.01 (0.12)
  Upper Leg Length(Thigh)-Knee to Heel Length Ratio | -0.01 (0.08) | 0.01 (0.07) | -0.09 (0.10) | -0.03 (0.08) | 0.01 (0.16) | -0.02 (0.11)
  Upper Leg Length (Thigh) to Tibial Length Ratio | 0.00 (0.12) | 0.02 (0.17) | -0.16 (0.24) | -0.10 (0.07) | 0.00 (0.29) | 0.04 (0.22)
  Arm Span to Standing Height Ratio: number analyzed (Participants) | 16 | 19 | 7 | 10 | 8 | 10
  Arm Span to Standing Height Ratio | 0.00 (0.02) | 0.00 (0.06) | 0.00 (0.02) | -0.01 (0.02) | -0.01 (0.04) | -0.02 (0.07)

8. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Week 52
Description: Body Mass Index (BMI): For height used for BMI calculation, participants aged < 24 months, body length takes precedence over standing height. Participants aged < 24 months at baseline and >= 24 months at Week 52, body length takes precedence.
Time Frame: Baseline to Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide | Cohort 3: Placebo | Cohort 3: Vosoritide
Number analyzed (Participants) | 16 | 19 | 7 | 12 | 8 | 11
kg/m^2 | 0.20 (1.34) | -0.45 (0.94) | 0.55 (1.17) | 0.08 (0.75) | 0.74 (1.70) | 0.94 (1.42)

9. Secondary Outcome: Change From Baseline in BMI Z-score at Week 52
Description: The body mass index (BMI) Z-score represents the participant's BMI converted to an age and sex appropriate standard deviation score (SDS) by comparison with an average stature reference population. The weight Z-score of 0 represents the mean BMI for age and sex of the reference population. A positive BMI Z-score means BMI is above the mean BMI for the average stature population of the same sex and age and a negative BMI Z-Score means BMI is below the mean BMI for the average stature population of the same sex and age.
  BMI Z-scores are derived only for participants aged 24 months or older, the change from baseline to Week 52 in BMI Z-score is summarized for Cohort 1 only as no participants in Cohort 2 or Cohort 3 were 24 months at baseline.
Time Frame: Baseline to Week 52
Population: FAS population.
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide
Number analyzed (Participants) | 16 | 19
Z-Score | -0.12 (0.48) | -0.18 (0.65)

10. Secondary Outcome: Change From Baseline in Weight Z-score at Week 52
Description: The weight Z-score represents the participant's weight converted to an age and sex appropriate standard deviation score (SDS) by comparison with an average stature reference population. The weight Z-score of 0 represents the mean weight for age and sex of the reference population. A positive weight Z-score means weight is above the mean weight for the average stature population of the same sex and age and a negative weight Z-Score means weight is below the mean weight for the average stature population of the same sex and age.
Time Frame: Baseline to Week 52
Population: FAS population
  Change from baseline was based on the subjects with available measurements at both time points. Baseline is defined as Day 1 or screening if a Day 1 measurement is not available
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide | Cohort 3: Placebo | Cohort 3: Vosoritide
Number analyzed (Participants) | 16 | 19 | 7 | 12 | 8 | 11
Z-score | 0.14 (0.44) | 0.14 (0.42) | 0.74 (0.82) | 0.70 (0.64) | -0.81 (0.49) | -0.66 (0.77)

11. Secondary Outcome: Change From Baseline in Infant Toddler Quality of Life (ITQoL) Scores at Week 52
Description: 97(ITQOL) item full-length version was used. For each concept, item responses are scored, summed, & transformed on a scale from 0(worst health) to 100(best health).
Time Frame: Baseline to Week 52
Population: FAS population.
  Change from baseline was based on the subjects with available measurements at both time points. Baseline is defined as Day 1 or screening if a Day 1 assessment is not available.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide | Cohort 3: Placebo | Cohort 3: Vosoritide
Number analyzed (Participants) | 14 | 17 | 7 | 12 | 8 | 10
Score on a scale
  Overall Health Score: number analyzed (Participants) | 12 | 15 | 5 | 10 | 6 | 10
  Overall Health Score | 3.75 (17.60) | 4.33 (15.10) | -5.00 (15.41) | -3.50 (14.15) | -5.00 (7.75) | 0.50 (13.01)
  Physical Abilities Score: number analyzed (Participants) | 14 | 17 | 7 | 12 | 7 | 6
  Physical Abilities Score | -6.01 (9.83) | 8.82 (23.06) | 3.36 (8.62) | 1.30 (16.05) | 2.35 (29.29) | -15.91 (22.74)
  Growth and Development Scores | 4.82 (11.62) | 4.34 (9.40) | -0.71 (8.75) | 1.46 (26.01) | 3.57 (6.35) | -3.50 (13.19)
  Pain Score | -1.19 (20.37) | -1.47 (18.22) | -1.19 (18.90) | -7.64 (27.63) | -4.69 (27.77) | 2.50 (22.58)
  Temperament and mood Score | 4.79 (9.60) | 0.54 (5.40) | 0.66 (7.18) | -0.49 (9.78) | -2.43 (6.76) | 4.62 (10.48)
  Global health perceptions score: number analyzed (Participants) | 13 | 17 | 7 | 12 | 8 | 9
  Global health perceptions score | -1.07 (15.43) | 2.24 (12.37) | -2.73 (11.29) | -4.55 (12.18) | -2.84 (13.62) | 0.50 (17.11)
  Parental impact emotional score | 2.04 (23.13) | -0.84 (8.89) | 0.51 (14.64) | -6.85 (11.94) | 9.82 (20.89) | -2.50 (19.05)
  Parental Impact Time Score | 9.52 (29.06) | 4.76 (10.78) | -8.05 (19.70) | -2.38 (35.61) | -10.7 (17.59) | 2.38 (14.93)
  Family Cohesion Score: number analyzed (Participants) | 14 | 16 | 7 | 12 | 8 | 10
  Family Cohesion Score | 1.79 (13.53) | -1.25 (10.72) | 0.00 (15.00) | -7.08 (28.08) | -3.13 (8.84) | -4.50 (15.54)

12. Secondary Outcome: Change From Baseline in ITQoL-Behavior Scores at Week 52
Description: 97(ITQOL) item full-length version was used. For each concept, item responses are scored, summed, & transformed on a scale from 0(worst health) to 100(best health).
  The number of subjects assessed in Cohort 3 Placebo is 0 as assessment was not done or overall score could not be derived because no more than half assessments were done at Screening/ baseline. Hence, Mean and Standard Deviation (SD) are not applicable.
  Note: For each variable, there are different numbers of individual questions. The variable can only be derived if at least half of the questions were completed.
Time Frame: Baseline to Week 52
Population: Full Analysis Set.
  Change from baseline was based on the subjects with available measurements at both time points. Baseline is defined as Day 1 or screening if a Day 1 assessment is not available.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Cohort 3 Placebo: Cohort 3 Placebo: Participants stratified by age 0 to < 6 months, received placebo single daily subcutaneous injection.
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide | Cohort 3: Vosoritide | Cohort 3 Placebo
Number analyzed (Participants) | 13 | 17 | 5 | 8 | 1 | 0
Score on a scale | 2.73 (23.36) | 0.37 (9.50) | 1.74 (13.60) | -3.39 (7.46) | 0.00 (NA) — As the number of subjects assessed in this category is only 1, Standard Deviation (SD) is not applicable. Hence SD values are proposed as NA. |

13. Secondary Outcome: Change From Baseline in ITQoL-Global Behavior Scores at Week 52
Description: 97(ITQOL) item full-length version was used. For each concept, item responses are scored, summed, & transformed on a scale from 0(worst health) to 100(best health). A higher score indicates better global behaviour.
  The number of subjects assessed in Cohort 3 Placebo is 0 as assessment was not done or overall score could not be derived because no more than half assessments were done at Screening/ baseline. Hence, Mean and Standard Deviation (SD) are not applicable.
  Note: For each variable, there are different numbers of individual questions. The variable can only be derived if at least half of the questions were completed.
Time Frame: Baseline to Week 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide | Cohort 3: Vosoritide | Cohort 3: Placebo
Number analyzed (Participants) | 13 | 17 | 5 | 9 | 1 | 0
Score on a scale | 1.15 (21.42) | 0.29 (18.58) | 3.00 (12.55) | -10.56 (21.71) | -15.00 (NA) — As the number of subjects assessed in this category is only 1, Standard Deviation (SD) is not applicable. Hence SD values are proposed as NA. |

14. Secondary Outcome: Change From Baseline in ITQoL-Getting On With Other Score at Week 52
Description: 97(ITQOL) item full-length version was used. For each concept, item responses are scored, summed, & transformed on a scale from 0(worst health) to 100(best health). A higher score indicates better global health perceptions.
  The number of subjects assessed in Cohort 3 Placebo and Cohort 3 vosoritide are 0 as assessment was not done or overall score could not be derived because no more than half assessments were done at Screening/baseline. Hence, Mean and Standard Deviation (SD) are not applicable.
  Note: For each variable, there are different numbers of individual questions. The variable can only be derived if at least half of the questions were completed.
Time Frame: Baseline to Week 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide | Cohort 3: Placebo | Cohort 3: Vosoritide
Number analyzed (Participants) | 12 | 17 | 5 | 8 | 0 | 0
Score on a scale | 7.78 (17.18) | 1.74 (8.88) | 2.33 (7.22) | 0.82 (5.35) |  |

15. Secondary Outcome: Change From Baseline in ITQoL-Health Score at Week 52
Description: 97(ITQOL) item full-length version was used. For each concept, item responses are scored, summed, & transformed on a scale from 0(worst health) to 100(best health). A higher score indicates better global change in health.
  The number of subjects assessed in Cohort 3 Placebo is 0 as assessment was not done or overall score could not be derived because no more than half assessments were done at Screening/ baseline. Hence, Mean and Standard Deviation (SD) are not applicable.
  Note: For each variable, there are different numbers of individual questions. The variable can only be derived if at least half of the questions were completed.
Time Frame: Baseline to Week 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide | Cohort 3: Vosoritide | Cohort 3: Placebo
Number analyzed (Participants) | 13 | 16 | 5 | 6 | 1 | 0
Score on a scale | 0.08 (0.64) | 0.13 (0.62) | -0.60 (1.34) | 0.33 (0.52) | 0.00 (NA) — As the number of subjects assessed in this category is only 1, standard deviation (SD) is not applicable. Hence SD value is proposed as NA. |

16. Secondary Outcome: Change From Baseline in Functional Independence Measure for Children (WeeFIM-II) Score at Week 52
Description: The Pediatric Functional Independence Measure-II (WeeFIM®-II) is designed to measure functional independence of children between the ages of 6 months & 18 yrs who have physical or general developmental limitations. The WeeFIM-II is comprised of 3 domains that are rated by clinicians based on information obtained from parents/caregivers (self-care [score range 8 to 56], mobility [score range 8 to 35], & cognition [score range 8 to 35]) & provides a total score between 18 (worst) & 126 (Best). Higher score reflects higher level of independence.
  Performance of a child on each of individual items within WeeFIM is assigned to one of seven levels on an ordinal scale that represent function from complete & modified independence (levels 7 & 6) without a helping person to modified & complete dependence (levels 5 to 1) with a helping person.
  Functional Independence Measure (Wee-FIM-II) is only validated in children ages 6 months to 18 yrs. Therefore results for Cohort 3 is not summarized.
Time Frame: Baseline to Week 52
Population: FAS population
  Change from baseline was based on the subjects with available measurements at both time points. Baseline is defined as Day 1 or screening if a Day 1 assessment is not available.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide
Number analyzed (Participants) | 14 | 19 | 6 | 11
Score on a scale
  WeeFIM-II Total Score | 11.2 (11.1) | 14.7 (17.3) | 16.2 (14.6) | 16.5 (28.1)
  WeeFIM : Self-Care Score | 6.4 (6.0) | 6.6 (7.2) | 3.7 (2.3) | 5.6 (14.1)
  WeeFIM: Mobility Score | 2.2 (3.4) | 4.5 (5.6) | 7.0 (7.5) | 6.7 (9.4)
  WeeFIM: Cognitive Score | 2.6 (4.0) | 3.6 (6.0) | 5.5 (7.6) | 4.2 (8.4)

17. Secondary Outcome: Change From Baseline in Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) Scores at Week 52
Description: BSID-III is performance-based clinician-reported outcome assessment for use in children from 1 to 42 months (1 month to 3.5 years). individually administered by the trained clinician to the participant/child
  Scales include Cognitive subscale, Receptive and Expressive subscales, and Gross and Fine Motor subscales. The two language scales make up a composite Language Scale score and the Gross and Fine Motor subscales yield a composite Motor Scale score. In addition, there is a Social-Emotional Scale and Adaptive Behavior Scale, which is a questionnaire read and completed by parent or caregiver. Scores range from 0 to 2, and indicate mastery (2), emerging (1) or zero (not present)
  Each (sub)scale yields a total raw score, standardized according to the participant's chronological age (scaled scores)
Time Frame: Baseline to Week 52
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide | Cohort 3: Placebo | Cohort 3: Vosoritide
Number analyzed (Participants) | 2 | 4 | 4 | 9 | 6 | 9
Score on a scale
  Motor Composite Score: number analyzed (Participants) | 2 | 4 | 4 | 9 | 5 | 8
  Motor Composite Score | -2.0 (5.7) | 4.8 (11.5) | 12.0 (17.5) | -2.3 (12.3) | 5.4 (22.2) | 11.1 (18.1)
  Cognitive scaled score: number analyzed (Participants) | 2 | 4 | 3 | 8 | 6 | 9
  Cognitive scaled score | -1.0 (2.8) | -0.5 (1.7) | 3.3 (4.9) | 0.6 (3.2) | 1.5 (1.9) | 2.1 (4.4)
  Cognitive composite score: number analyzed (Participants) | 2 | 4 | 3 | 8 | 6 | 9
  Cognitive composite score | -5.0 (14.1) | -2.5 (8.7) | 16.7 (24.7) | 3.1 (16.0) | 7.5 (9.4) | 10.6 (22.1)
  Receptive communication language scaled score: number analyzed (Participants) | 2 | 4 | 3 | 9 | 5 | 9
  Receptive communication language scaled score | -1.0 (0.0) | -1.8 (2.5) | 3.3 (4.0) | 1.0 (1.2) | -3.0 (2.1) | 0.7 (5.2)
  Expressive communication language scaled score: number analyzed (Participants) | 2 | 4 | 4 | 8 | 5 | 8
  Expressive communication language scaled score | 2.5 (0.7) | 0.3 (1.3) | 2.8 (2.9) | -0.1 (2.2) | -1.8 (1.6) | -0.1 (3.3)
  Language sum of scaled score | 1.5 (0.7) | -1.5 (3.3) | 6.0 (5.2) | 1.8 (4.0) | -7.3 (6.4) | -0.3 (6.6)
  Language composite score: number analyzed (Participants) | 2 | 4 | 4 | 9 | 5 | 9
  Language composite score | 4.5 (2.1) | -4.5 (9.9) | 17.8 (15.2) | 5.3 (12.1) | -13.4 (5.8) | -0.9 (19.5)
  Fine motor scaled score: number analyzed (Participants) | 2 | 4 | 4 | 9 | 5 | 8
  Fine motor scaled score | -0.5 (3.5) | 0.0 (2.9) | 1.5 (3.3) | -2.1 (2.5) | 2.2 (4.8) | 2.6 (2.7)
  Gross motor scaled score: number analyzed (Participants) | 2 | 4 | 4 | 9 | 5 | 9
  Gross motor scaled score | 0.0 (5.7) | 1.0 (0.8) | 2.8 (3.2) | 1.3 (2.8) | -0.2 (3.1) | 0.1 (3.0)

18. Secondary Outcome: Change From Baseline in Child Behaviour Checklist (CBCL) at Week 52
Description: The CBCL is used as a screening tool for emotional or behavioral problems, measuring initial behavior severity, tracking changes in behavioral problems over the course of treatment, and treatment planning. The CBCL 1.5-5 years old consists of 100 questions, scored on a three-point Likert scale (0=Not True (as far as you know), 1= Somewhat or Sometimes True, 2=Very True or Often True). The scores for each individual question within a domain are summed to give a domain score. The CBCL uses a normative sample to create standard scores, which are scaled so that 50 is average with a standard deviation of 10, where higher scores indicate more emotional or behavioral issues.
  CBCL was waived for children < 18 months old. Therefore results for Cohort 3 is not summarized.
Time Frame: Baseline to Week 52
Population: Safety population
  Change from baseline was based on the subjects with available measurements at both time points. Baseline is defined as Day 1 or screening if a Day 1 assessment is not available.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide
Number analyzed (Participants) | 15 | 18 | 4 | 5
Score on a scale
  CBCL Pre-School : Emotionally Reactive Total | -0.2 (1.5) | 0.1 (1.4) | 1.0 (2.0) | 1.0 (3.9)
  CBCL Pre-School : Anxious/Depressed Total | 0.3 (1.7) | 0.2 (1.4) | 0.0 (2.2) | 0.8 (3.1)
  CBCL Pre-School : Withdrawn Total | -0.6 (1.7) | 0.6 (1.5) | 0.8 (2.2) | -0.2 (1.6)
  CBCL Pre-School : Somatic Complaints Total | 0.1 (1.7) | 0.3 (1.0) | 0.5 (1.0) | 1.8 (4.1)
  CBCL Pre-School : Sleep Problems Total | -0.3 (3.2) | 0.1 (1.9) | -0.3 (1.7) | 1.4 (4.3)
  CBCL Pre-School : Attention Problems Total | -0.1 (1.9) | -0.1 (1.6) | -0.3 (1.0) | -0.2 (2.0)
  CBCL Pre-School : Aggressive Behavior Total | -1.1 (2.4) | 0.3 (4.1) | -0.8 (1.5) | -0.4 (2.7)
  CBCL Pre-School : Total Problems Total | -3.0 (13.0) | 2.8 (11.7) | -2.3 (6.0) | 3.6 (23.2)

19. Secondary Outcome: Change From Baseline in Bilateral X-rays of Lower Extremities at Week 52
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 40 | 27
cm
  Left Femur Length: number analyzed (Participants) | 17 | 14
  Left Femur Length | 2.29 (0.58) | 2.01 (0.62)
  Right Femur Length: number analyzed (Participants) | 17 | 14
  Right Femur Length | 2.35 (0.49) | 2.20 (0.73)
  Left Fibula Length | 2.00 (0.61) | 1.97 (0.69)
  Right Fibula Length: number analyzed (Participants) | 39 | 27
  Right Fibula Length | 2.00 (0.64) | 1.89 (0.75)
  Left Tibia Length | 1.92 (0.55) | 1.69 (0.70)
  Right Tibia Length: number analyzed (Participants) | 39 | 27
  Right Tibia Length | 1.96 (0.57) | 1.68 (0.77)
  Left Distance Between Ankle Joint and Distal Growth Plate of Fibula: number analyzed (Participants) | 38 | 26
  Left Distance Between Ankle Joint and Distal Growth Plate of Fibula | -0.02 (0.23) | 0.07 (0.23)
  Right Distance Between Ankle Joint and Distal Growth Plate of Fibula: number analyzed (Participants) | 37 | 26
  Right Distance Between Ankle Joint and Distal Growth Plate of Fibula | -0.05 (0.23) | 0.05 (0.22)
  Left Lower Extremity: number analyzed (Participants) | 18 | 14
  Left Lower Extremity | 6.02 (6.67) | 3.87 (1.56)
  Right Lower Extremity: number analyzed (Participants) | 18 | 14
  Right Lower Extremity | 6.08 (6.54) | 4.26 (1.85)

20. Secondary Outcome: Change From Baseline in Bilateral X-rays of Left/Right Tibia Bowing Angle at Week 52
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 39 | 27
Degrees
  Left Tibia Bowing Angle | -0.97 (5.88) | 1.07 (5.38)
  Right Tibia Bowing Angle: number analyzed (Participants) | 38 | 27
  Right Tibia Bowing Angle | -2.34 (5.37) | -0.93 (5.54)

21. Secondary Outcome: Change From Baseline in Bilateral X-rays of Left Femur Length (cm) to Tibia Length (cm) Ratio and Right Femur Length (cm) to Tibia Length (cm) Ratio at Week 52
Time Frame: Baseline to Week 52 End point timeframe:
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 17 | 14
Ratio
  Left Femur Length (cm) to Tibia Length (cm) Ratio | -0.03 (0.06) | -0.05 (0.05)
  Right Femur Length (cm) to Tibia Length (cm) Ratio | -0.05 (0.06) | -0.02 (0.03)

22. Secondary Outcome: Change From Baseline in Bilateral X-rays of Left Tibia Length (cm) to Fibula Length (cm) Ratio & Right Tibia Length (cm) to Fibula Length (cm) Ratio at Week 52
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 40 | 27
Ratio
  Left Tibia Length (cm) to Fibula Length (cm) Ratio | -0.02 (0.04) | -0.04 (0.04)
  Right Tibia Length (cm) to Fibula Length(cm) Ratio: number analyzed (Participants) | 39 | 27
  Right Tibia Length (cm) to Fibula Length(cm) Ratio | -0.02 (0.05) | -0.03 (0.04)

23. Secondary Outcome: Change From Baseline in X-ray of Lumbar Spine Vertebral Ratios at Week 52
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 40 | 27
Ratio
  Anterior Height to Medial Height Ratio (L1): number analyzed (Participants) | 30 | 23
  Anterior Height to Medial Height Ratio (L1) | -0.04 (0.16) | -0.04 (0.20)
  Anterior Height to Medial Height Ratio (L2): number analyzed (Participants) | 23 | 13
  Anterior Height to Medial Height Ratio (L2) | -0.06 (0.16) | -0.07 (0.16)
  Anterior Height to Medial Height Ratio (L3): number analyzed (Participants) | 19 | 11
  Anterior Height to Medial Height Ratio (L3) | -0.02 (0.19) | 0.04 (0.09)
  Anterior Height to Medial Height Ratio (L4): number analyzed (Participants) | 26 | 15
  Anterior Height to Medial Height Ratio (L4) | 0.02 (0.12) | -0.01 (0.11)
  Anterior Height to Medial Height Ratio (L5): number analyzed (Participants) | 27 | 12
  Anterior Height to Medial Height Ratio (L5) | -0.02 (0.15) | 0.04 (0.17)
  Anterior Height to Posterior Height Ratio (L1) | -0.03 (0.13) | -0.08 (0.17)
  Anterior Height to Posterior Height Ratio (L2) | -0.02 (0.13) | -0.03 (0.12)
  Anterior Height to Posterior Height Ratio (L3) | -0.01 (0.16) | 0.04 (0.12)
  Anterior Height to Posterior Height Ratio (L4) | 0.03 (0.11) | 0.02 (0.13)
  Anterior Height to Posterior Height Ratio (L5) | 0.01 (0.13) | 0.02 (0.15)
  Medial Height to Posterior Height Ratio (L1): number analyzed (Participants) | 30 | 23
  Medial Height to Posterior Height Ratio (L1) | -0.01 (0.15) | -0.04 (0.12)
  Medial Height to Posterior Height Ratio (L2): number analyzed (Participants) | 23 | 13
  Medial Height to Posterior Height Ratio (L2) | 0.05 (0.11) | 0.03 (0.09)
  Medial Height to Posterior Height Ratio (L3): number analyzed (Participants) | 19 | 11
  Medial Height to Posterior Height Ratio (L3) | -0.02 (0.10) | -0.02 (0.10)
  Medial Height to Posterior Height Ratio (L4): number analyzed (Participants) | 26 | 15
  Medial Height to Posterior Height Ratio (L4) | -0.03 (0.13) | 0.04 (0.10)
  Medial Height to Posterior Height Ratio (L5): number analyzed (Participants) | 27 | 12
  Medial Height to Posterior Height Ratio (L5) | 0.02 (0.16) | -0.04 (0.21)

24. Secondary Outcome: Change From Baseline in X-ray of Lumbar Spine Transverse Diameter at Week 52
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 40 | 27
cm
  Transverse Diameter (L1) | 0.12 (0.17) | 0.12 (0.11)
  Transverse Diameter (L2) | 0.12 (0.16) | 0.09 (0.13)
  Transverse Diameter (L3) | 0.08 (0.15) | 0.09 (0.12)
  Transverse Diameter (L4) | 0.09 (0.13) | 0.06 (0.11)
  Transverse Diameter (L5) | 0.10 (0.13) | 0.05 (0.14)

25. Secondary Outcome: Change From Baseline in X-ray of Lumbar Spine Sagittal Width and Week 52
Description: Baseline is defined as Day 1 or screening if a Day 1 assessment is not available.
Time Frame: Baseline to Week 52
Population: Safety population
  Change from baseline was based on subjects with available measurements at both time points. Overall no. of participants analyzed (N) is greater than no. analyzed for Placebo, as different participants missed for different variables (Ex:1 subject missed sagittal width L1,L2,L3, 1 subject missed sagittal width L5 & 1 subject missed sagittal width L4 & L5. Therefore, n for sagittal width L1,L2,L3,L4 & L5 are 26,26,26,26,25 respectively but the overall number of subjects is 27)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 34 | 27
cm
  Sagittal Width (L1): number analyzed (Participants) | 34 | 26
  Sagittal Width (L1) | 0.07 (0.26) | 0.00 (0.22)
  Sagittal Width (L2): number analyzed (Participants) | 34 | 26
  Sagittal Width (L2) | 0.05 (0.18) | 0.01 (0.18)
  Sagittal Width (L3): number analyzed (Participants) | 34 | 26
  Sagittal Width (L3) | 0.08 (0.20) | 0.04 (0.19)
  Sagittal Width (L4): number analyzed (Participants) | 34 | 26
  Sagittal Width (L4) | 0.16 (0.24) | 0.03 (0.16)
  Sagittal Width (L5): number analyzed (Participants) | 31 | 25
  Sagittal Width (L5) | 0.13 (0.34) | 0.06 (0.26)

26. Secondary Outcome: Change From Baseline in X-ray of Lumbar Spine Angles at Week 52
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 40 | 27
Degree
  Sacral Tilt | 10.6 (13.2) | 5.7 (15.9)
  Lordosis Angle | 12.5 (17.4) | 8.4 (14.2)
  Kyphosis Angle: number analyzed (Participants) | 39 | 27
  Kyphosis Angle | -2.2 (13.9) | -2.1 (10.3)

27. Secondary Outcome: Changes From Baseline in X-ray of Lumbar Spine Angle Changes: Number of Participants With an Increase in Lumbar Spine Angle at Week 52
Description: Percentages were calculated using the total number of subjects in the safety population (N for each treatment group) as the denominator.
  All increases are comparing results at Week 52 relative to the baseline assessment.
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Number; unit: Number of participants
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 37 | 21
Number of participants
  Increase in sacral tilt (deg) >=5 to <10 | 3 | 6
  Increase in sacral tilt (deg) >=10 | 24 | 10
  Increase in lordosis angle (deg) >=5 to <10 | 5 | 1
  Increase in lordosis angle (deg) >=10 | 19 | 14
  Increase in kyphosis angle (deg) >=5 to <10 | 3 | 2
  Increase in kyphosis angle (deg) >=10 | 9 | 4

28. Secondary Outcome: MRI Parameter: Change From Baseline to Week 52 for Volume of Face, Sinus, Calvarium, Whole Brain Total Volume, Ventricles Total Volume.
Time Frame: Baseline to Week 52
Population: Safety population
  Change from baseline and percent change from baseline are based on the subjects with available measurements at both time points. Baseline is defined as Day 1 or screening if a Day 1 assessment is not available.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 35 | 25
cm^3
  Volume of Face: number analyzed (Participants) | 30 | 21
  Volume of Face | 80.527 (59.211) | 78.107 (33.369)
  Volume of Sinus: number analyzed (Participants) | 35 | 24
  Volume of Sinus | 2.362 (3.578) | 1.195 (3.769)
  Volume of Calvarium: number analyzed (Participants) | 34 | 24
  Volume of Calvarium | 213.075 (202.415) | 183.427 (183.210)
  Whole Brain Total Volume: number analyzed (Participants) | 34 | 24
  Whole Brain Total Volume | 175.399 (158.088) | 146.247 (115.274)
  Ventricles Total Volume: number analyzed (Participants) | 34 | 25
  Ventricles Total Volume | 11.394 (20.416) | 8.515 (16.325)

29. Secondary Outcome: MRI Parameter: Percentage Change From Baseline to Week 52 for Volume of Face, Sinus, Calvarium, Whole Brain Total Volume, Ventricles Total Volume.
Time Frame: Baseline to Week 52
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 35 | 25
percent change
  Volume of Face: number analyzed (Participants) | 30 | 21
  Volume of Face | 20.79 (18.46) | 19.18 (12.22)
  Volume of sinus: number analyzed (Participants) | 35 | 24
  Volume of sinus | 72.33 (100.93) | 81.97 (169.74)
  Volume of Calvarium: number analyzed (Participants) | 34 | 24
  Volume of Calvarium | 19.41 (21.73) | 16.50 (19.82)
  Whole Brain Total Volume: number analyzed (Participants) | 34 | 24
  Whole Brain Total Volume | 20.58 (21.29) | 16.89 (17.22)
  Ventricles Total Volume: number analyzed (Participants) | 34 | 25
  Ventricles Total Volume | 33.44 (52.69) | 30.85 (50.65)

30. Secondary Outcome: MRI Parameter: Change From Baseline to Week 52 for Area of Foramen Magnum & Area of Spinal Cord at the Foramen Magnum Level
Time Frame: Baseline to Week 52
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 35 | 25
cm^2
  Area of Foramen Magnum | 0.021 (0.342) | 0.060 (0.203)
  Area of Spinal Cord at the Foramen Magnum Level | 0.011 (0.197) | 0.072 (0.163)

31. Secondary Outcome: MRI Parameter: Percentage Change From Baseline to Week 52 for Area of Foramen Magnum & Area of Spinal Cord at the Foramen Magnum Level
Time Frame: Baseline to Week 52
Population: Safety Population.
  Change from baseline and percent change from baseline are based on the subjects with available measurements at both time points. Baseline is defined as Day 1 or screening if a Day 1 assessment is not available.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 35 | 25
Percent change
  Area of Foramen Magnum | 9.19 (47.36) | 7.50 (19.88)
  Area of spinal cord at the foramen magnum level | 7.51 (33.14) | 19.60 (44.26)

32. Secondary Outcome: MRI Parameter: Change From Baseline to Week 52 for Ratio of Face Volume to Calvarium, Ratio of Area of Spinal Cord to Foramen Magnum, Ratio of Face Volume to Sinus
Time Frame: Baseline to Week 52
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 35 | 25
Ratio
  Ratio of face volume to calvarium: number analyzed (Participants) | 29 | 20
  Ratio of face volume to calvarium | 0.002 (0.031) | 0.003 (0.033)
  Ratio of area of spinal cord to foramen magnum | 0.005 (0.120) | 0.037 (0.100)
  Ratio of face volume to sinus: number analyzed (Participants) | 30 | 21
  Ratio of face volume to sinus | -6.798 (175.646) | 14.505 (284.950)

33. Secondary Outcome: MRI Parameter: Percentage Change From Baseline to Week 52 for Ratio of Face Volume to Calvarium, Ratio of Area of Spinal Cord to Foramen Magnum, Ratio of Face Volume to Sinus
Time Frame: Baseline to Week 52
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 35 | 25
Percent change
  Ratio of Face Volume to Calvarium: number analyzed (Participants) | 29 | 20
  Ratio of Face Volume to Calvarium | 0.78 (9.06) | 1.31 (10.07)
  Ratio of Area of Spinal Cord to Foramen Magnum | 2.86 (23.40) | 9.50 (22.68)
  Ratio of face volume to sinus: number analyzed (Participants) | 30 | 21
  Ratio of face volume to sinus | -5.37 (60.83) | 92.24 (341.33)

34. Secondary Outcome: Dual X Ray Absorptiometry (DEXA) Parameter: Change From Baseline to Week 52 for Whole Body Less Head Bone Mineral Content (BMC)
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: gm
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 26 | 20
gm
  GE - Lunar Prodigy: Whole Body Less Head BMC: number analyzed (Participants) | 8 | 12
  GE - Lunar Prodigy: Whole Body Less Head BMC | 55.87 (14.68) | 50.26 (17.44)
  Hologic Discovery Horizon Whole Body Less Head BMC: number analyzed (Participants) | 18 | 8
  Hologic Discovery Horizon Whole Body Less Head BMC | 44.61 (12.62) | 47.19 (12.55)

35. Secondary Outcome: DEXA Parameter: Change From Baseline to Week 52 of Whole Body Less Head Bone Mineral Density (BMD)
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 26 | 20
g/cm^2
  GE - Lunar Prodigy Whole Body Less Head BMD: number analyzed (Participants) | 8 | 12
  GE - Lunar Prodigy Whole Body Less Head BMD | 0.04 (0.02) | 0.05 (0.03)
  Hologic Discovery Horizon Whole Body Less Head BMD: number analyzed (Participants) | 18 | 8
  Hologic Discovery Horizon Whole Body Less Head BMD | 0.03 (0.01) | 0.04 (0.02)

36. Secondary Outcome: DEXA Parameter: Change From Baseline to Week 52 of Whole Body BMC
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: gm
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 26 | 20
gm
  GE - Lunar Prodigy Whole Body BMC: number analyzed (Participants) | 8 | 12
  GE - Lunar Prodigy Whole Body BMC | 96.85 (39.82) | 98.99 (32.45)
  Hologic - Discovery Horizon Whole Body BMC: number analyzed (Participants) | 18 | 8
  Hologic - Discovery Horizon Whole Body BMC | 87.97 (32.35) | 101.33 (33.34)

37. Secondary Outcome: DEXA Parameter: Change From Baseline to Week 52 of Lumbar Spine BMC
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: gm
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 36 | 23
gm
  GE - Lunar Prodigy Lumbar Spine BMC: number analyzed (Participants) | 9 | 10
  GE - Lunar Prodigy Lumbar Spine BMC | 2.73 (0.83) | 2.09 (0.97)
  Hologic - Discovery Horizon Lumbar Spine BMC: number analyzed (Participants) | 27 | 13
  Hologic - Discovery Horizon Lumbar Spine BMC | 2.19 (0.68) | 1.94 (0.72)

38. Secondary Outcome: DEXA Parameter: Change From Baseline to Week 52 of Whole Body BMD
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 26 | 20
g/cm^2
  GE - Lunar Prodigy Whole Body BMD: number analyzed (Participants) | 8 | 12
  GE - Lunar Prodigy Whole Body BMD | 0.06 (0.06) | 0.07 (0.04)
  Hologic - Discovery Horizon Whole Body BMD: number analyzed (Participants) | 18 | 8
  Hologic - Discovery Horizon Whole Body BMD | 0.05 (0.02) | 0.07 (0.03)

39. Secondary Outcome: DEXA Parameter: Change From Baseline to Week 52 of Lumbar Spine BMD
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 36 | 23
g/cm^2
  GE - Lunar Prodigy Lumbar Spine BMD: number analyzed (Participants) | 9 | 10
  GE - Lunar Prodigy Lumbar Spine BMD | 0.07 (0.04) | 0.05 (0.03)
  Hologic - Discovery Horizon Lumbar Spine BMD: number analyzed (Participants) | 27 | 13
  Hologic - Discovery Horizon Lumbar Spine BMD | 0.05 (0.03) | 0.06 (0.04)

40. Secondary Outcome: Change From Baseline to Week 52 in Whole Body BMD Z-score
Description: Hologic - Discovery Horizon Whole Body BMD Z-Score.
  Change in whole body bone mineral density (BMD) Z-score from baseline at 52 weeks indicates whether there has been a positive or negative change in BMD using a z-score generated by converting the participants BMD to an age and sex appropriate standard deviation score (SDS) by comparison with an average stature reference population. A whole body BMD Z-score <-2 SD can indicate low bone density in children. The Whole Body BMD (bone mineral density) z-score compares the BMD to the average bone density of people of the same age, and sex as a comparator. A Z-score less than 0 means that the participant has a lower BMD than people in the same age and sex group, and could indicate a risk of osteopenia or osteoporosis.
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 6 | 4
Z-score | -0.20 (0.35) | 0.30 (0.47)

41. Secondary Outcome: Change From Baseline to Week 52 in Lumbar Spine BMD Z-Score
Description: Hologic - Discovery Horizon Lumbar Spine BMD Z-Score
  Change in lumbar spine bone mineral density (BMD) Z-score from baseline at 52 weeks indicates whether there has been a positive or negative change in BMD using a z-score generated by converting the participants lumbar spine BMD to an age and sex appropriate standard deviation score (SDS) by comparison with an average stature reference population. A BMD Z-score <-2 SD can indicate low bone density in the lumbar spine in children. The Lumbar Spine BMD (bone mineral density) z-score compares the BMD in the lumbar spine to the average spinal bone density of people of the same age, and sex as a comparator. A Z-score less than 0 means that the participant has a lower BMD than people in the same age and sex group, and could indicate a risk of osteopenia or osteoporosis of the spine.
Time Frame: Baseline to Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 7 | 4
Z-score | 0.17 (0.24) | 0.03 (0.45)

42. Secondary Outcome: Immunogenicity: Number of Participants With Incidence of Antibody Positivity at Scheduled Visits
Description: Number of participants with Incidence of Antibody Positivity at Scheduled Visits for : total antibody (TAb), Neutralizing antibodies (NAb), atrial natriuretic peptide (ANP), B-type Natriuretic Peptide (BNP) & C-type natriuretic peptide (CNP).
  TAb Titer Positive, NAb Titer Positive, ANP Reactivity Positive, BNP Reactivity Positive & CNP Reactivity Positive.
  Day 1 is the baseline assessment result taken prior to first dose of study drug.
  Ever Positive = the number of participants with at least one positive sample result.
Time Frame: At Day 1, Week 3, Week 13, Week 26, Week 52, & Ever Positive.
Population: FAS population
Measure: Number; unit: participants
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 43 | 32
participants
  TAb Titer Positive: Day 1: number analyzed (Participants) | 37 | 31
  TAb Titer Positive: Day 1 | 0 | 0
  TAb Titer Positive: Week 3: number analyzed (Participants) | 22 | 20
  TAb Titer Positive: Week 3 | 0 | 0
  TAb Titer Positive: Week 13: number analyzed (Participants) | 37 | 29
  TAb Titer Positive: Week 13 | 0 | 0
  TAb Titer Positive: Week 26: number analyzed (Participants) | 36 | 29
  TAb Titer Positive: Week 26 | 2 | 0
  TAb Titer Positive: Week 52: number analyzed (Participants) | 33 | 28
  TAb Titer Positive: Week 52 | 8 | 0
  TAb Titer Ever Positive | 8 | 0
  NAb Titer Positive: Day 1: number analyzed (Participants) | 37 | 31
  NAb Titer Positive: Day 1 | 0 | 0
  NAb Titer Positive: Week 3: number analyzed (Participants) | 22 | 20
  NAb Titer Positive: Week 3 | 0 | 0
  NAb Titer Positive: Week 13: number analyzed (Participants) | 37 | 29
  NAb Titer Positive: Week 13 | 0 | 0
  NAb Titer Positive: Week 26: number analyzed (Participants) | 36 | 29
  NAb Titer Positive: Week 26 | 0 | 0
  NAb Titer Positive: Week 52: number analyzed (Participants) | 33 | 28
  NAb Titer Positive: Week 52 | 0 | 0
  NAb Titer Ever Positive | 0 | 0
  ANP Reactivity Positive: Day 1: number analyzed (Participants) | 37 | 31
  ANP Reactivity Positive: Day 1 | 3 | 5
  ANP Reactivity Positive: Week 3: number analyzed (Participants) | 22 | 20
  ANP Reactivity Positive: Week 3 | 0 | 0
  ANP Reactivity Positive: Week 13: number analyzed (Participants) | 37 | 29
  ANP Reactivity Positive: Week 13 | 1 | 0
  ANP Reactivity Positive: Week 26: number analyzed (Participants) | 36 | 29
  ANP Reactivity Positive: Week 26 | 6 | 0
  ANP Reactivity Positive: Week 52: number analyzed (Participants) | 33 | 28
  ANP Reactivity Positive: Week 52 | 11 | 0
  ANP Reactivity Ever Positive | 12 | 0
  BNP Reactivity Positive: Day 1: number analyzed (Participants) | 37 | 31
  BNP Reactivity Positive: Day 1 | 0 | 3
  BNP Reactivity Positive: Week 3: number analyzed (Participants) | 22 | 20
  BNP Reactivity Positive: Week 3 | 0 | 0
  BNP Reactivity Positive: Week 13: number analyzed (Participants) | 37 | 29
  BNP Reactivity Positive: Week 13 | 2 | 0
  BNP Reactivity Positive: Week 26: number analyzed (Participants) | 36 | 29
  BNP Reactivity Positive: Week 26 | 3 | 0
  BNP Reactivity Positive: Week 52: number analyzed (Participants) | 33 | 28
  BNP Reactivity Positive: Week 52 | 2 | 0
  BNP Reactivity Ever Positive | 3 | 0
  CNP Reactivity Positive: Day 1: number analyzed (Participants) | 37 | 31
  CNP Reactivity Positive: Day 1 | 0 | 1
  CNP Reactivity Positive: Week 3: number analyzed (Participants) | 22 | 20
  CNP Reactivity Positive: Week 3 | 0 | 0
  CNP Reactivity Positive: Week 13: number analyzed (Participants) | 37 | 29
  CNP Reactivity Positive: Week 13 | 1 | 0
  CNP Reactivity Positive: Week 26: number analyzed (Participants) | 36 | 29
  CNP Reactivity Positive: Week 26 | 2 | 0
  CNP Reactivity Positive: Week 52: number analyzed (Participants) | 33 | 28
  CNP Reactivity Positive: Week 52 | 4 | 0
  CNP Reactivity Ever Positive | 4 | 0

43. Secondary Outcome: Biomarker: Bone Specific Alkaline Phosphatase (BSAP) Overtime
Time Frame: At Baseline, Day 8, Week 6, Week 20, & Week 39.
Population: Safety population
  Change from baseline and percent change from baseline are based on the subjects with available measurements at both time points. Baseline is the last measurement prior to the initiation of study drug.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 43 | 32
U/L
  BSAP: Baseline | 140.28 (183.23) | 113.43 (33.56)
  BSAP: Day 8: number analyzed (Participants) | 42 | 27
  BSAP: Day 8 | 122.32 (99.09) | 104.12 (29.12)
  BSAP: Change from baseline to Day 8: number analyzed (Participants) | 42 | 27
  BSAP: Change from baseline to Day 8 | -19.39 (202.90) | -7.67 (17.53)
  BSAP: Week 6: number analyzed (Participants) | 41 | 29
  BSAP: Week 6 | 130.38 (140.08) | 109.46 (29.04)
  BSAP: Change from baseline to Week 6: number analyzed (Participants) | 41 | 29
  BSAP: Change from baseline to Week 6 | 2.63 (218.60) | -6.17 (24.32)
  BSAP: Week 20: number analyzed (Participants) | 40 | 28
  BSAP: Week 20 | 109.67 (30.88) | 104.46 (29.69)
  BSAP: Change from baseline to Week 20: number analyzed (Participants) | 40 | 28
  BSAP: Change from baseline to Week 20 | -7.21 (96.94) | -11.32 (18.19)
  BSAP: Week 39: number analyzed (Participants) | 34 | 24
  BSAP: Week 39 | 108.49 (32.02) | 208.13 (363.56)
  BSAP: Change from baseline to Week 39: number analyzed (Participants) | 34 | 24
  BSAP: Change from baseline to Week 39 | -12.21 (105.04) | 95.41 (352.78)

44. Secondary Outcome: Biomarker: Type II Collagen C-Telopeptides Normalized for Creatinine (CTX-II)
Time Frame: Baseline to Week 52.
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: ng/ mmol Cr
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 31 | 24
ng/ mmol Cr | -9364.7 (65244.1) | -7607.6 (54614.9)

45. Secondary Outcome: Biomarker: Plasma Cyclic Guanosine Monophosphate (cGMP) Change From Pre-Dose to Maximum Post-Dose at Week 52
Time Frame: Week 52 Pre-Dose to Week 52 Maximum Post-Dose.
Population: Safety population. Change from baseline and percent change from baseline are based on the subjects with available measurements at both time points. Baseline is the last measurement prior to the initiation of study drug.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 33 | 21
nM | 39.079 (25.706) | 9.460 (26.307)

46. Secondary Outcome: Biomarker: Bone and Collagen Metabolism Biomarker Over Time-CNP Col X BM
Description: Laboratory results up to 30 days after study drug discontinuation were included.
  Baseline is the last measurement prior to the initiation of study drug.
Time Frame: At Baseline, Day 8, Week 6, Week 20, & Week 39.
Population: Safety Population.
  Change from baseline was based on subjects with available measurements at both timepoints.Overall no. of participants analyzed(N) is greater than no. analyzed for All Vosoritide, as different participants missed for different timepoints(Ex:1 of 42 participants who were part of CNP Col X BM:Baseline was not present in 42 participants who participated in CNP Col X BM:Day 8.Therefore, n for CNP Col X BM:Baseline & CNP Col X BM:Day 8 are 42 however, overall no of subjects,N=43)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | All Vosoritide | Placebo
Number analyzed (Participants) | 43 | 32
pg/mL
  CNP Col X BM: Baseline: number analyzed (Participants) | 42 | 32
  CNP Col X BM: Baseline | 9833.8 (3444.7) | 9555.0 (4016.7)
  CNP Col X BM: Day 8: number analyzed (Participants) | 42 | 24
  CNP Col X BM: Day 8 | 12093.8 (4443.8) | 10017.5 (3831.2)
  CNP Col X BM: Change from baseline to Day 8: number analyzed (Participants) | 41 | 24
  CNP Col X BM: Change from baseline to Day 8 | 2139.5 (3871.9) | 1391.3 (3354.2)
  CNP Col X BM: Week 6: number analyzed (Participants) | 41 | 29
  CNP Col X BM: Week 6 | 13456.3 (4763.3) | 9464.8 (4243.3)
  CNP Col X BM: Change from baseline to Week 6: number analyzed (Participants) | 40 | 29
  CNP Col X BM: Change from baseline to Week 6 | 3400.3 (4554.6) | 200.3 (3867.5)
  CNP Col X BM: Week 20: number analyzed (Participants) | 42 | 29
  CNP Col X BM: Week 20 | 12833.3 (4581.9) | 12064.8 (5277.3)
  CNP Col X BM: Change from baseline to Week 20: number analyzed (Participants) | 41 | 29
  CNP Col X BM: Change from baseline to Week 20 | 2928.0 (4385.9) | 2435.5 (4666.9)
  CNP Col X BM: Week 39: number analyzed (Participants) | 33 | 22
  CNP Col X BM: Week 39 | 12249.7 (5056.5) | 9932.7 (4004.4)
  CNP Col X BM: Change from baseline to Week 39: number analyzed (Participants) | 32 | 22
  CNP Col X BM: Change from baseline to Week 39 | 2362.8 (5752.9) | 946.4 (3490.1)

47. Secondary Outcome: Change in Sleep Study Indices at Week 52
Description: Sleep-testing device was used to assess presence & severity of sleep-disordered breathing by measurement of blood oxygen(O2)saturation,pulse rate,& airflow during overnight monitoring
  Episodes(Epi) of sleep apnea variables summarized as: Number(No.)of epi of apnea/hr(AI);No.of epi of hypopnea/hr(HI);No.of epi of obstructive apnea hypopneas/hr(AHI);No.of epi of obstructive apneas/hr(Obstructive Apnea Index);No.of epi of central apneas/hr(CAI);No.of desaturations/hr >=3%
  AHI is a marker of obstructive sleep apnea (OSA), scored as No.of apnea or hypopnea epi/hr, with AHI <=1/hr normal, 1< AHI<=5 mild,5< AHI <=10 moderate,& AHI>10/hr severe OSA. CAI reflects cervical cord compression at cervical-medullary junction, & is No. of epi of a pause in ventilation with no associated respiratory effort, with> 5 epi/hr abnormal.O2 desaturation index measures average No. of desaturation epi/hr, defined as decrease in O2 saturation of >=3% for at least 10sec, with(<8/hr normal & >=8/hr abnormal
Time Frame: Baseline to Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Events per hour
Arm/Group | Cohort 1: Placebo | Cohort 1: Vosoritide | Cohort 2: Placebo | Cohort 2: Vosoritide | Cohort 3: Placebo | Cohort 3: Vosoritide
Number analyzed (Participants) | 14 | 16 | 5 | 9 | 7 | 10
Events per hour
  Apnea Hypopnea Index (AHI) | -0.54 (2.70) | -1.45 (4.63) | 1.06 (4.80) | -0.72 (1.41) | 1.89 (6.31) | -0.94 (2.78)
  Apnea Index (AI) | -1.07 (2.12) | -0.83 (1.93) | 0.40 (2.34) | -0.71 (1.61) | -1.09 (1.22) | -0.36 (2.54)
  Central Apnea Index (CAI) | -1.26 (2.66) | -0.74 (1.86) | -0.28 (0.89) | -0.71 (1.61) | -1.00 (0.97) | 0.50 (0.92)
  Hypopnea Index (HI) | 0.52 (1.35) | -0.61 (3.63) | 0.66 (2.53) | -0.01 (1.32) | 2.97 (5.45) | -0.56 (0.54)
  Desaturation per Hour >=3% | -0.41 (1.51) | -1.24 (3.98) | 0.98 (3.60) | -0.69 (1.30) | 1.71 (6.63) | -0.93 (2.60)
  Obstructive Index | 0.19 (0.73) | -0.09 (0.45) | 0.68 (1.52) | -0.01 (0.08) | -0.07 (0.64) | -0.86 (2.08)

48. Secondary Outcome: PK Parameter: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-∞) at Day1, Week 13, Week 26, Week 39, & Week 52
Description: Vosoritide concentrations at 5-, 15- and 30-minute post-dose for one participant on Day 1 were not available, hence PK parameters for this participant were excluded from summary statistics.
  PK parameters for another participant on Day 1 obtained from extrapolation. AUC0-∞ excluded from summary statistics. PK parameters are not available for this participant at Week 13 due to unsuccessful venipuncture, and Week 26 as post-dose PK samples were not collected.
Time Frame: At Day1, Week 13, Week 26, Week 39, & Week 52.
Population: Pharmacokinetics (PK) Population includes all sentinel and randomized participants in the safety population who have at least one evaluable PK concentration.
Measure: Mean (Standard Deviation); unit: min*pg/ml
Arm/Group | All Vosoritide
Number analyzed (Participants) | 43
min*pg/ml
  Cohort 1 15 μg/kg/day: Day 01: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Day 01 | 149000 (98000)
  Cohort 1 15 μg/kg/day: Week 13: number analyzed (Participants) | 15
  Cohort 1 15 μg/kg/day: Week 13 | 197000 (144000)
  Cohort 1 15 μg/kg/day: Week 26: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 26 | 306000 (252000)
  Cohort 1 15 μg/kg/day: Week 39: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 39 | 284000 (137000)
  Cohort 1 15 μg/kg/day: Week 52: number analyzed (Participants) | 15
  Cohort 1 15 μg/kg/day: Week 52 | 303000 (208000)
  Cohort 2 15 μg/kg/day: Day 01: number analyzed (Participants) | 1
  Cohort 2 15 μg/kg/day: Day 01 | 102000 (NA) — As the number of subjects assessed in this category is only 1, Standard Deviation (SD) is not applicable. Hence SD value is proposed as NA.
  Cohort 2 15 μg/kg/day: Week 13: number analyzed (Participants) | 1
  Cohort 2 15 μg/kg/day: Week 13 | 74500 (NA) — As the number of subjects assessed in this category is only 1, Standard Deviation (SD) is not applicable. Hence SD value is proposed as NA.
  Cohort 2 15 μg/kg/day: Week 26: number analyzed (Participants) | 4
  Cohort 2 15 μg/kg/day: Week 26 | 233000 (132000)
  Cohort 2 15 μg/kg/day: Week 39: number analyzed (Participants) | 4
  Cohort 2 15 μg/kg/day: Week 39 | 204000 (39700)
  Cohort 2 15 μg/kg/day: Week 52: number analyzed (Participants) | 3
  Cohort 2 15 μg/kg/day: Week 52 | 137000 (48900)
  Cohort 2 30 μg/kg/day: Day 01: number analyzed (Participants) | 7
  Cohort 2 30 μg/kg/day: Day 01 | 557000 (278000)
  Cohort 2 30 μg/kg/day: Week 13: number analyzed (Participants) | 6
  Cohort 2 30 μg/kg/day: Week 13 | 670000 (312000)
  Cohort 2 30 μg/kg/day: Week 26: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 26 | 429000 (163000)
  Cohort 2 30 μg/kg/day: Week 39: number analyzed (Participants) | 2
  Cohort 2 30 μg/kg/day: Week 39 | 387000 (53800)
  Cohort 2 30 μg/kg/day: Week 52: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 52 | 768000 (391000)
  Cohort 3 30 μg/kg/day: Day 01: number analyzed (Participants) | 8
  Cohort 3 30 μg/kg/day: Day 01 | 353000 (133000)
  Cohort 3 30 μg/kg/day: Week 13: number analyzed (Participants) | 6
  Cohort 3 30 μg/kg/day: Week 13 | 382000 (268000)
  Cohort 3 30 μg/kg/day: Week 26: number analyzed (Participants) | 6
  Cohort 3 30 μg/kg/day: Week 26 | 305000 (82100)
  Cohort 3 30 μg/kg/day: Week 39: number analyzed (Participants) | 3
  Cohort 3 30 μg/kg/day: Week 39 | 575000 (455000)
  Cohort 3 30 μg/kg/day: Week 52: number analyzed (Participants) | 7
  Cohort 3 30 μg/kg/day: Week 52 | 622000 (455000)

49. Secondary Outcome: PK Parameter: Area Under the Plasma Concentration-time Curve From Time 0 to Nominal 120 Minutes Postdose (AUC 0- 120 Min) at Day 01, Week 13, Week 26, Week 39, & Week 52
Time Frame: At Day 01, Week 13, Week 26, Week 39, & Week 52
Population: PK Population
Measure: Mean (Standard Deviation); unit: min*pg/ml
Arm/Group | All Vosoritide
Number analyzed (Participants) | 43
min*pg/ml
  Cohort 1 15 μg/kg/day: Day 01: number analyzed (Participants) | 18
  Cohort 1 15 μg/kg/day: Day 01 | 134000 (96500)
  Cohort 1 15 μg/kg/day: Week 13: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 13 | 183000 (126000)
  Cohort 1 15 μg/kg/day: Week 26: number analyzed (Participants) | 17
  Cohort 1 15 μg/kg/day: Week 26 | 283000 (222000)
  Cohort 1 15 μg/kg/day: Week 39: number analyzed (Participants) | 19
  Cohort 1 15 μg/kg/day: Week 39 | 257000 (132000)
  Cohort 1 15 μg/kg/day: Week 52: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 52 | 260000 (172000)
  Cohort 2 15 μg/kg/day: Day 01: number analyzed (Participants) | 3
  Cohort 2 15 μg/kg/day: Day 01 | 83100 (48300)
  Cohort 2 15 μg/kg/day: Week 13: number analyzed (Participants) | 2
  Cohort 2 15 μg/kg/day: Week 13 | 115000 (59300)
  Cohort 2 15 μg/kg/day: Week 26: number analyzed (Participants) | 5
  Cohort 2 15 μg/kg/day: Week 26 | 197000 (121000)
  Cohort 2 15 μg/kg/day: Week 39: number analyzed (Participants) | 5
  Cohort 2 15 μg/kg/day: Week 39 | 166000 (81000)
  Cohort 2 15 μg/kg/day: Week 52: number analyzed (Participants) | 5
  Cohort 2 15 μg/kg/day: Week 52 | 125000 (76700)
  Cohort 2 30 μg/kg/day: Day 01: number analyzed (Participants) | 7
  Cohort 2 30 μg/kg/day: Day 01 | 525000 (251000)
  Cohort 2 30 μg/kg/day: Week 13: number analyzed (Participants) | 8
  Cohort 2 30 μg/kg/day: Week 13 | 642000 (353000)
  Cohort 2 30 μg/kg/day: Week 26: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 26 | 408000 (148000)
  Cohort 2 30 μg/kg/day: Week 39: number analyzed (Participants) | 2
  Cohort 2 30 μg/kg/day: Week 39 | 365000 (44700)
  Cohort 2 30 μg/kg/day: Week 52: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 52 | 670000 (335000)
  Cohort 3 30 μg/kg/day: Day 01: number analyzed (Participants) | 11
  Cohort 3 30 μg/kg/day: Day 01 | 312000 (119000)
  Cohort 3 30 μg/kg/day: Week 13: number analyzed (Participants) | 7
  Cohort 3 30 μg/kg/day: Week 13 | 342000 (245000)
  Cohort 3 30 μg/kg/day: Week 26: number analyzed (Participants) | 6
  Cohort 3 30 μg/kg/day: Week 26 | 300000 (79100)
  Cohort 3 30 μg/kg/day: Week 39: number analyzed (Participants) | 4
  Cohort 3 30 μg/kg/day: Week 39 | 591000 (359000)
  Cohort 3 30 μg/kg/day: Week 52: number analyzed (Participants) | 8
  Cohort 3 30 μg/kg/day: Week 52 | 558000 (400000)

50. Secondary Outcome: PK Parameter: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of Last Measurable Concentration (AUC0-t) at Day 01, Week 13, Week 26, Week 39, & Week 52
Time Frame: At Day 01, Week 13, Week 26, Week 39, & Week 52
Population: PK Population
Measure: Mean (Standard Deviation); unit: min*pg/ml
Arm/Group | All Vosoritide
Number analyzed (Participants) | 43
min*pg/ml
  Cohort 1 15 μg/kg/day: Day 01: number analyzed (Participants) | 18
  Cohort 1 15 μg/kg/day: Day 01 | 132000 (97300)
  Cohort 1 15 μg/kg/day: Week 13: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 13 | 182000 (127000)
  Cohort 1 15 μg/kg/day: Week 26: number analyzed (Participants) | 17
  Cohort 1 15 μg/kg/day: Week 26 | 282000 (222000)
  Cohort 1 15 μg/kg/day: Week 39: number analyzed (Participants) | 19
  Cohort 1 15 μg/kg/day: Week 39 | 256000 (132000)
  Cohort 1 15 μg/kg/day: Week 52: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 52 | 258000 (169000)
  Cohort 2 15 μg/kg/day: Day 01: number analyzed (Participants) | 3
  Cohort 2 15 μg/kg/day: Day 01 | 65900 (33600)
  Cohort 2 15 μg/kg/day: Week 13: number analyzed (Participants) | 2
  Cohort 2 15 μg/kg/day: Week 13 | 112000 (62900)
  Cohort 2 15 μg/kg/day: Week 26: number analyzed (Participants) | 5
  Cohort 2 15 μg/kg/day: Week 26 | 196000 (121000)
  Cohort 2 15 μg/kg/day: Week 39: number analyzed (Participants) | 5
  Cohort 2 15 μg/kg/day: Week 39 | 165000 (82400)
  Cohort 2 15 μg/kg/day: Week 52: number analyzed (Participants) | 5
  Cohort 2 15 μg/kg/day: Week 52 | 122000 (75700)
  Cohort 2 30 μg/kg/day: Day 01: number analyzed (Participants) | 7
  Cohort 2 30 μg/kg/day: Day 01 | 547000 (279000)
  Cohort 2 30 μg/kg/day: Week 13: number analyzed (Participants) | 8
  Cohort 2 30 μg/kg/day: Week 13 | 645000 (357000)
  Cohort 2 30 μg/kg/day: Week 26: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 26 | 407000 (148000)
  Cohort 2 30 μg/kg/day: Week 39: number analyzed (Participants) | 2
  Cohort 2 30 μg/kg/day: Week 39 | 365000 (44300)
  Cohort 2 30 μg/kg/day: Week 52: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 52 | 672000 (334000)
  Cohort 3 30 μg/kg/day: Day 01: number analyzed (Participants) | 11
  Cohort 3 30 μg/kg/day: Day 01 | 323000 (129000)
  Cohort 3 30 μg/kg/day: Week 13: number analyzed (Participants) | 7
  Cohort 3 30 μg/kg/day: Week 13 | 340000 (244000)
  Cohort 3 30 μg/kg/day: Week 26: number analyzed (Participants) | 6
  Cohort 3 30 μg/kg/day: Week 26 | 297000 (80700)
  Cohort 3 30 μg/kg/day: Week 39: number analyzed (Participants) | 4
  Cohort 3 30 μg/kg/day: Week 39 | 567000 (361000)
  Cohort 3 30 μg/kg/day: Week 52: number analyzed (Participants) | 8
  Cohort 3 30 μg/kg/day: Week 52 | 557000 (401000)

51. Secondary Outcome: PK Parameter: Maximum Observed Plasma Concentration (Cmax) at Day 01, Week 13, Week 26, Week 39, & Week 52
Time Frame: At Day 01, Week 13, Week 26, Week 39, & Week 52
Population: PK Population
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | All Vosoritide
Number analyzed (Participants) | 43
pg/ml
  Cohort 1 15 μg/kg/day: Day 01: number analyzed (Participants) | 18
  Cohort 1 15 μg/kg/day: Day 01 | 4430 (3670)
  Cohort 1 15 μg/kg/day: Week 13: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 13 | 4350 (1670)
  Cohort 1 15 μg/kg/day: Week 26: number analyzed (Participants) | 17
  Cohort 1 15 μg/kg/day: Week 26 | 5850 (3260)
  Cohort 1 15 μg/kg/day: Week 39: number analyzed (Participants) | 19
  Cohort 1 15 μg/kg/day: Week 39 | 5600 (2200)
  Cohort 1 15 μg/kg/day: Week 52: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 52 | 5640 (2740)
  Cohort 2 15 μg/kg/day: Day 01: number analyzed (Participants) | 3
  Cohort 2 15 μg/kg/day: Day 01 | 2840 (1230)
  Cohort 2 15 μg/kg/day: Week 13: number analyzed (Participants) | 2
  Cohort 2 15 μg/kg/day: Week 13 | 5970 (2390)
  Cohort 2 15 μg/kg/day: Week 26: number analyzed (Participants) | 5
  Cohort 2 15 μg/kg/day: Week 26 | 6800 (3360)
  Cohort 2 15 μg/kg/day: Week 39: number analyzed (Participants) | 5
  Cohort 2 15 μg/kg/day: Week 39 | 4600 (2150)
  Cohort 2 15 μg/kg/day: Week 52: number analyzed (Participants) | 5
  Cohort 2 15 μg/kg/day: Week 52 | 3870 (2120)
  Cohort 2 30 μg/kg/day: Day 01: number analyzed (Participants) | 7
  Cohort 2 30 μg/kg/day: Day 01 | 14500 (5950)
  Cohort 2 30 μg/kg/day: Week 13: number analyzed (Participants) | 8
  Cohort 2 30 μg/kg/day: Week 13 | 13400 (6070)
  Cohort 2 30 μg/kg/day: Week 26: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 26 | 10100 (2970)
  Cohort 2 30 μg/kg/day: Week 39: number analyzed (Participants) | 2
  Cohort 2 30 μg/kg/day: Week 39 | 6980 (1140)
  Cohort 2 30 μg/kg/day: Week 52: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 52 | 12900 (6260)
  Cohort 3 30 μg/kg/day: Day 01: number analyzed (Participants) | 11
  Cohort 3 30 μg/kg/day: Day 01 | 13400 (5710)
  Cohort 3 30 μg/kg/day: Week 13: number analyzed (Participants) | 7
  Cohort 3 30 μg/kg/day: Week 13 | 10500 (6850)
  Cohort 3 30 μg/kg/day: Week 26: number analyzed (Participants) | 6
  Cohort 3 30 μg/kg/day: Week 26 | 11500 (4290)
  Cohort 3 30 μg/kg/day: Week 39: number analyzed (Participants) | 4
  Cohort 3 30 μg/kg/day: Week 39 | 18400 (11900)
  Cohort 3 30 μg/kg/day: Week 52: number analyzed (Participants) | 8
  Cohort 3 30 μg/kg/day: Week 52 | 13500 (6770)

52. Secondary Outcome: PK Parameter: Time to Reach Maximum Concentration (Tmax) at Day 01, Week 13, Week 26, Week 39, & Week 52
Time Frame: At Day 01, Week 13, Week 26, Week 39, & Week 52.
Population: PK Population
Measure: Mean (Standard Deviation); unit: min
Arm/Group | All Vosoritide
Number analyzed (Participants) | 43
min
  Cohort 1 15 μg/kg/day: Day 01: number analyzed (Participants) | 18
  Cohort 1 15 μg/kg/day: Day 01 | 13.1 (6.33)
  Cohort 1 15 μg/kg/day: Week 13: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 13 | 14.3 (5.5)
  Cohort 1 15 μg/kg/day: Week 26: number analyzed (Participants) | 17
  Cohort 1 15 μg/kg/day: Week 26 | 16.1 (8.69)
  Cohort 1 15 μg/kg/day: Week 39: number analyzed (Participants) | 19
  Cohort 1 15 μg/kg/day: Week 39 | 17.4 (11.9)
  Cohort 1 15 μg/kg/day: Week 52: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 52 | 16.1 (6.27)
  Cohort 2 15 μg/kg/day: Day 01: number analyzed (Participants) | 3
  Cohort 2 15 μg/kg/day: Day 01 | 11.3 (6.35)
  Cohort 2 15 μg/kg/day: Week 13: number analyzed (Participants) | 2
  Cohort 2 15 μg/kg/day: Week 13 | 6 (1.41)
  Cohort 2 15 μg/kg/day: Week 26: number analyzed (Participants) | 5
  Cohort 2 15 μg/kg/day: Week 26 | 10.8 (5.5)
  Cohort 2 15 μg/kg/day: Week 39: number analyzed (Participants) | 5
  Cohort 2 15 μg/kg/day: Week 39 | 15.4 (11.6)
  Cohort 2 15 μg/kg/day: Week 52: number analyzed (Participants) | 5
  Cohort 2 15 μg/kg/day: Week 52 | 14.2 (5.76)
  Cohort 2 30 μg/kg/day: Day 01: number analyzed (Participants) | 7
  Cohort 2 30 μg/kg/day: Day 01 | 12.9 (9.1)
  Cohort 2 30 μg/kg/day: Week 13: number analyzed (Participants) | 8
  Cohort 2 30 μg/kg/day: Week 13 | 14 (8.42)
  Cohort 2 30 μg/kg/day: Week 26: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 26 | 12 (5.2)
  Cohort 2 30 μg/kg/day: Week 39: number analyzed (Participants) | 2
  Cohort 2 30 μg/kg/day: Week 39 | 15 (0)
  Cohort 2 30 μg/kg/day: Week 52: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 52 | 14.3 (1.53)
  Cohort 3 30 μg/kg/day: Day 01: number analyzed (Participants) | 11
  Cohort 3 30 μg/kg/day: Day 01 | 7.36 (3.53)
  Cohort 3 30 μg/kg/day: Week 13: number analyzed (Participants) | 7
  Cohort 3 30 μg/kg/day: Week 13 | 9.43 (5.22)
  Cohort 3 30 μg/kg/day: Week 26: number analyzed (Participants) | 6
  Cohort 3 30 μg/kg/day: Week 26 | 9 (4.69)
  Cohort 3 30 μg/kg/day: Week 39: number analyzed (Participants) | 4
  Cohort 3 30 μg/kg/day: Week 39 | 11.3 (3.59)
  Cohort 3 30 μg/kg/day: Week 52: number analyzed (Participants) | 8
  Cohort 3 30 μg/kg/day: Week 52 | 14.5 (3.51)

53. Secondary Outcome: PK Parameter: Apparent Clearance (CL/F) at Day 01, Week 13, Week 26, Week 39, & Week 52
Description: Vosoritide concentrations at 5-, 15- and 30-minute post-dose for one participant on Day 1 were not available, hence PK parameters for this participant were excluded from summary statistics.
  PK parameters for another participant on Day 1 obtained from extrapolation. AUC0-∞, CL/F, V/F and t1/2 excluded from summary statistics. PK parameters are not available for this participant at Week 13 due to unsuccessful venipuncture, and Week 26 as post-dose PK samples were not collected.
Time Frame: At Day 01, Week 13, Week 26, Week 39, & Week 52.
Population: PK Population
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | All Vosoritide
Number analyzed (Participants) | 43
ml/min/kg
  Cohort 1 15 μg/kg/day: Day 01: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Day 01 | 134 (59.8)
  Cohort 1 15 μg/kg/day: Week 13: number analyzed (Participants) | 15
  Cohort 1 15 μg/kg/day: Week 13 | 111 (58.5)
  Cohort 1 15 μg/kg/day: Week 26: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 26 | 79.8 (48.3)
  Cohort 1 15 μg/kg/day: Week 39: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 39 | 65.3 (32.7)
  Cohort 1 15 μg/kg/day: Week 52: number analyzed (Participants) | 15
  Cohort 1 15 μg/kg/day: Week 52 | 69 (41.2)
  Cohort 2 15 μg/kg/day: Day 1: number analyzed (Participants) | 1
  Cohort 2 15 μg/kg/day: Day 1 | 147 (NA) — As the number of subjects assessed in this category is only 1, Standard Deviation (SD) is not applicable. Hence SD value is proposed as NA.
  Cohort 2 15 μg/kg/day: Week 13: number analyzed (Participants) | 1
  Cohort 2 15 μg/kg/day: Week 13 | 201 (NA) — As the number of subjects assessed in this category is only 1, Standard Deviation (SD) is not applicable. Hence SD value is proposed as NA.
  Cohort 2 15 μg/kg/day: Week 26: number analyzed (Participants) | 4
  Cohort 2 15 μg/kg/day: Week 26 | 79.5 (38.4)
  Cohort 2 15 μg/kg/day: Week 39: number analyzed (Participants) | 4
  Cohort 2 15 μg/kg/day: Week 39 | 75.5 (14.8)
  Cohort 2 15 μg/kg/day: Week 52: number analyzed (Participants) | 3
  Cohort 2 15 μg/kg/day: Week 52 | 122 (52.5)
  Cohort 2 30 μg/kg/day: Day 01: number analyzed (Participants) | 7
  Cohort 2 30 μg/kg/day: Day 01 | 65.9 (31.6)
  Cohort 2 30 μg/kg/day: Week 13: number analyzed (Participants) | 6
  Cohort 2 30 μg/kg/day: Week 13 | 58.7 (40.4)
  Cohort 2 30 μg/kg/day: Week 26: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 26 | 79.4 (37.7)
  Cohort 2 30 μg/kg/day: Week 39: number analyzed (Participants) | 2
  Cohort 2 30 μg/kg/day: Week 39 | 78.3 (10.9)
  Cohort 2 30 μg/kg/day: Week 52: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 52 | 49.7 (32)
  Cohort 3 30 μg/kg/day: Day 01: number analyzed (Participants) | 8
  Cohort 3 30 μg/kg/day: Day 01 | 95.9 (34)
  Cohort 3 30 μg/kg/day: Week 13: number analyzed (Participants) | 6
  Cohort 3 30 μg/kg/day: Week 13 | 115 (78.1)
  Cohort 3 30 μg/kg/day: Week 26: number analyzed (Participants) | 6
  Cohort 3 30 μg/kg/day: Week 26 | 104 (23.2)
  Cohort 3 30 μg/kg/day: Week 39: number analyzed (Participants) | 3
  Cohort 3 30 μg/kg/day: Week 39 | 73.6 (41.6)
  Cohort 3 30 μg/kg/day: Week 52: number analyzed (Participants) | 7
  Cohort 3 30 μg/kg/day: Week 52 | 76.5 (49.8)

54. Secondary Outcome: PK Parameter: Apparent Volume of Distribution (Vz/F) at Day 01, Week 13, Week 26, Week 39, & Week 52
Description: Vosoritide concentrations at 5-, 15- and 30-minute post-dose for one participant on Day 1 were not available, hence PK parameters for this participant were excluded from summary statistics.
  PK parameters for another participant on Day 1 obtained from extrapolation. V/F excluded from summary statistics. PK parameters are not available for this participant at Week 13 due to unsuccessful venipuncture, and Week 26 as post-dose PK samples were not collected.
Time Frame: At Day 01, Week 13, Week 26, Week 39, & Week 52.
Population: PK Population
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | All Vosoritide
Number analyzed (Participants) | 43
ml/kg
  Cohort 1 15 μg/kg/day: Day 01: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Day 01 | 4070 (2310)
  Cohort 1 15 μg/kg/day: Week 13: number analyzed (Participants) | 15
  Cohort 1 15 μg/kg/day: Week 13 | 3990 (2960)
  Cohort 1 15 μg/kg/day: Week 26: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 26 | 3400 (2520)
  Cohort 1 15 μg/kg/day: Week 39: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 39 | 2330 (1150)
  Cohort 1 15 μg/kg/day: Week 52: number analyzed (Participants) | 15
  Cohort 1 15 μg/kg/day: Week 52 | 2660 (1420)
  Cohort 2 15 μg/kg/day: Day 01: number analyzed (Participants) | 1
  Cohort 2 15 μg/kg/day: Day 01 | 5550 (NA) — As the number of subjects assessed in this category is only 1, Standard Deviation (SD) is not applicable. Hence SD value is proposed as NA.
  Cohort 2 15 μg/kg/day: Week 13: number analyzed (Participants) | 1
  Cohort 2 15 μg/kg/day: Week 13 | 7810 (NA) — As the number of subjects assessed in this category is only 1, Standard Deviation (SD) is not applicable. Hence SD value is proposed as NA.
  Cohort 2 15 μg/kg/day: Week 26: number analyzed (Participants) | 4
  Cohort 2 15 μg/kg/day: Week 26 | 3890 (2880)
  Cohort 2 15 μg/kg/day: Week 39: number analyzed (Participants) | 4
  Cohort 2 15 μg/kg/day: Week 39 | 2250 (284)
  Cohort 2 15 μg/kg/day: Week 52: number analyzed (Participants) | 3
  Cohort 2 15 μg/kg/day: Week 52 | 3770 (1410)
  Cohort 2 30 μg/kg/day: Day 01: number analyzed (Participants) | 7
  Cohort 2 30 μg/kg/day: Day 01 | 3190 (1790)
  Cohort 2 30 μg/kg/day: Week 13: number analyzed (Participants) | 6
  Cohort 2 30 μg/kg/day: Week 13 | 2090 (1360)
  Cohort 2 30 μg/kg/day: Week 26: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 26 | 1960 (829)
  Cohort 2 30 μg/kg/day: Week 39: number analyzed (Participants) | 2
  Cohort 2 30 μg/kg/day: Week 39 | 2920 (205)
  Cohort 2 30 μg/kg/day: Week 52: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 52 | 3040 (2630)
  Cohort 3 30 μg/kg/day: Day 01: number analyzed (Participants) | 8
  Cohort 3 30 μg/kg/day: Day 01 | 5240 (1890)
  Cohort 3 30 μg/kg/day: Week 13: number analyzed (Participants) | 6
  Cohort 3 30 μg/kg/day: Week 13 | 4260 (2960)
  Cohort 3 30 μg/kg/day: Week 26: number analyzed (Participants) | 6
  Cohort 3 30 μg/kg/day: Week 26 | 2750 (710)
  Cohort 3 30 μg/kg/day: Week 39: number analyzed (Participants) | 3
  Cohort 3 30 μg/kg/day: Week 39 | 2200 (951)
  Cohort 3 30 μg/kg/day: Week 52: number analyzed (Participants) | 7
  Cohort 3 30 μg/kg/day: Week 52 | 2620 (1950)

55. Secondary Outcome: PK Parameter: Elimination Half-life (t1/2) at Day 01, Week 13, Week 26, Week 39, & Week 52
Description: as for outcome 53
Time Frame: At Day 01, Week 13, Week 26, Week 39, & Week 52.
Population: PK Population
Measure: Mean (Standard Deviation); unit: min
Arm/Group | All Vosoritide
Number analyzed (Participants) | 43
min
  Cohort 1 15 μg/kg/day: Day 01: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Day 01 | 21.7 (7.99)
  Cohort 1 15 μg/kg/day: Week 13: number analyzed (Participants) | 15
  Cohort 1 15 μg/kg/day: Week 13 | 25.4 (10.7)
  Cohort 1 15 μg/kg/day: Week 26: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 26 | 29.2 (7.06)
  Cohort 1 15 μg/kg/day: Week 39: number analyzed (Participants) | 16
  Cohort 1 15 μg/kg/day: Week 39 | 25.7 (7.82)
  Cohort 1 15 μg/kg/day: Week 52: number analyzed (Participants) | 15
  Cohort 1 15 μg/kg/day: Week 52 | 29 (9.12)
  Cohort 2 15 μg/kg/day: Day 01: number analyzed (Participants) | 1
  Cohort 2 15 μg/kg/day: Day 01 | 26.1 (NA) — As the number of subjects assessed in this category is only 1, Standard Deviation (SD) is not applicable. Hence SD value is proposed as NA.
  Cohort 2 15 μg/kg/day: Week 13: number analyzed (Participants) | 1
  Cohort 2 15 μg/kg/day: Week 13 | 26.9 (NA) — As the number of subjects assessed in this category is only 1, Standard Deviation (SD) is not applicable. Hence SD value is proposed as NA.
  Cohort 2 15 μg/kg/day: Week 26: number analyzed (Participants) | 4
  Cohort 2 15 μg/kg/day: Week 26 | 32.7 (9.62)
  Cohort 2 15 μg/kg/day: Week 39: number analyzed (Participants) | 4
  Cohort 2 15 μg/kg/day: Week 39 | 20.9 (2.18)
  Cohort 2 15 μg/kg/day: Week 52: number analyzed (Participants) | 3
  Cohort 2 15 μg/kg/day: Week 52 | 24 (12.8)
  Cohort 2 30 μg/kg/day: Day 01: number analyzed (Participants) | 7
  Cohort 2 30 μg/kg/day: Day 01 | 33.3 (8.41)
  Cohort 2 30 μg/kg/day: Week 13: number analyzed (Participants) | 6
  Cohort 2 30 μg/kg/day: Week 13 | 25.6 (3.59)
  Cohort 2 30 μg/kg/day: Week 26: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 26 | 21 (13.1)
  Cohort 2 30 μg/kg/day: Week 39: number analyzed (Participants) | 2
  Cohort 2 30 μg/kg/day: Week 39 | 26.2 (5.46)
  Cohort 2 30 μg/kg/day: Week 52: number analyzed (Participants) | 3
  Cohort 2 30 μg/kg/day: Week 52 | 40.1 (15.2)
  Cohort 3 30 μg/kg/day: Day 01: number analyzed (Participants) | 8
  Cohort 3 30 μg/kg/day: Day 01 | 41.1 (18.8)
  Cohort 3 30 μg/kg/day: Week 13: number analyzed (Participants) | 6
  Cohort 3 30 μg/kg/day: Week 13 | 26.2 (7.1)
  Cohort 3 30 μg/kg/day: Week 26: number analyzed (Participants) | 6
  Cohort 3 30 μg/kg/day: Week 26 | 19.2 (6.14)
  Cohort 3 30 μg/kg/day: Week 39: number analyzed (Participants) | 3
  Cohort 3 30 μg/kg/day: Week 39 | 22.7 (5.36)
  Cohort 3 30 μg/kg/day: Week 52: number analyzed (Participants) | 7
  Cohort 3 30 μg/kg/day: Week 52 | 24.3 (6.58)

ADVERSE EVENTS:
Time Frame: Up to Week 56 Safety Follow-Up.
Description: The Safety Population was a subset of the FAS who received at least one dose of vosoritide or placebo in the study.
  The safety data is presented for the overall vosoritide and placebo cohort. The doses for each of the cohorts were selected such that the exposure to vosoritide, based on pharmacokinetic parameters, was comparable across all 3 cohorts.
Groups:
- Vosoritide: All Vosoritide : 11 sentinel + 32 randomized participants who received vosoritide 15 µg/kg/day or 30 µg/kg/day, single daily subcutaneous injection.
Arm/Group | Placebo | Vosoritide
All-Cause Mortality (participants affected / at risk) | 0/32 | 1/43
Serious Adverse Events (participants affected / at risk) | 6/32 | 3/43
Other Adverse Events (participants affected / at risk) | 32/32 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | Vosoritide (N=43)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Autism spectrum disorde (Psychiatric disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Sudden infant death syndrome (General disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | Vosoritide (N=43)
Rhinitis (Infections and infestations) | 0 (0) | 4 (8)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (3) | 4 (4)
Viral infection (Infections and infestations) | 4 (8) | 8 (28)
Injection site reaction (General disorders) | 13 (154) | 34 (3057)
Injection site erythema (General disorders) | 13 (1738) | 33 (5100)
Injection site swelling (General disorders) | 2 (3) | 8 (36)
Injection site induration (General disorders) | 0 (0) | 5 (14)
Injection site urticaria (General disorders) | 1 (1) | 6 (22)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (4) | 5 (7)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 7 (9)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 6 (7)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT03583697/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT03583697/SAP_001.pdf